## Statistical Analysis Plan (SAP) – Primary Analysis (APHAB)

**Project:** Evaluation of Unilateral vs Bilateral Hearing Aids for the Treatment of Age-related Hearing Loss **IRB Number:** Pro00106077 Investigator(s): Sherri Smith, AuD, PhD Biostatistician(s): **Original Creation Date:** 09.21.2021 Version Date: 11.13.2024 ☐ All statistical analyses included in an abstract or manuscript should **Investigator Agreement** reflect the work of the biostatistician(s) listed on this SAP. No changes or additional analyses should be made to the results or findings without discussing with the project biostatistician(s). ☐ All biostatisticians on this SAP should be given sufficient time to review the full presentation, abstract, manuscript, or grant and be included as co-authors on any abstract or manuscript resulting from the analyses. ☐ If substantial additional analysis is necessary or the aims of the project change, a new SAP will need to be developed. ☐ Publications resulting from this SAP are supported in part by the Duke CTSA and must cite grant number UL1TR002553 and be submitted to PubMed Central. □ I have reviewed the SAP and understand that any changes must be documented. Acknowledged by: Click or tap here to enter text. Date: Click or tap to enter a date. **Activity Log** 10.07.2021 Moved 6 month APHAB outcomes to separate SAP and edited based on feedback/comments in the 09.21.2021 SBP SAP. 11.01.2021 Added written models 01.20.2022 Edited document based on discussions 07.20.2022 Stratified Table 1 by randomization 11.17.2022 Added additional details to variables 12.15.2022 Edited based on discussions 06.28.2023 Refined ITT language 05.31.2024 Updated audiogram data information 07.11.2024 Added specific subgroup analysis (mild vs moderate) 09.30.2024 Added APHAB subscale change scores, specified primary analysis as "completers" analysis, changed benefit scores to change scores (3m-baseline), updated variable names, added information about adjusted models/subgroup models 10.28.2024 Added ineligible (missing) definition to binary APHAB change score in Section 3.2, date of data lock

NCT04739436 Page 1

| 11.13.2024 Moved tables to different order, removed tables for |
|------------------------------------------------------------------------|
| analyses we are not doing/created a subsection describing which |
| analyses we are not doing, updated heterogeneity of treatment effects |
| to only mention variables of interest, added variables of interest for |
| multiple imputation |

| Acronyms | АРНАВ | Abbreviated Profile of Hearing Aid Benefit |
|----------|----------|--------------------------------------------|
| | MoCA | Montreal Cognitive Assessment |
| | EC scale | Ease of Communication |
| | BN scale | Background Noise |
| | RV scale | Reverberation |
| | AV scale | Aversiveness |

# 1 Study Overview

Background/Introduction: The overall goal of the project is to determine the benefit of unilateral or bilateral hearing aid fittings in adults with mild-to-moderate age-related hearing loss. This will address the lack of high-quality evidence supporting bilateral hearing aids over unilateral hearing aids. This project will use a randomized controlled trial with two treatment arms: a bilateral hearing aid fitting group and a unilateral hearing aid fitting group.

#### 1.1 Primary Aims

• Compare the APHAB change scores between the two arms (bilateral hearing aid and unilateral hearing aid) at the end of month 3. The primary hypothesis is that bilateral hearing aids are superior to the unilateral hearing aids with respect to the overall patient-reported benefit.

#### 1.2 Secondary Aims

- Compare the APHAB change scores between the two arms at the end of month 3 while adjusting for covariates
- Compare the APHAB change scores between the two arms at the end of month 3 with subgroup analyses
- Sensitivity analysis with missing data
- Analyze APHAB binary response at 3 months
- Create descriptives for the 4 APHAB subscales in unaided (baseline) and aided conditions (3 month) for each arm

# 2 Study Population

### 2.1 Inclusion Criteria

- 50+ years of age
- Mild to moderate, symmetrical SNHL (symmetrical: < 20 dB between ears on average from 500-4000 Hz)
- Open-mindedness to unilateral or bilateral amplification
- No prior hearing aid experience
- Adequate literacy to complete questionnaires
- Willing to purchase study-specific hearing aid(s)

### 2.2 Exclusion Criteria

- Concerns for middle ear pathology
- Concerns for retrocochlear pathology
- Severe tinnitus as the reason for seeking amplification
- Co-morbid condition that would interfere with study (e.g., dementia, blindness, neurologic pathology)
- History of fluctuating hearing loss

### 2.3 Data Acquisition

Fill in all relevant information:

| Study design | Randomized controlled trial with 2 arms (bilateral |
|---|---|
| | hearing aid, unilateral hearing aid) |
| | Note: Randomization was stratified by clinical site. |
| Data source/how the data were collected | Screening information pulled from EHR data |
| | Baseline surveys captured via in-person interview and |
| | recorded in REDCap |
| Contact information for team member | All data access is through |
| responsible for data | . Questions on data validity |
| collection/acquisition | will go to PI: Sherri Smith (Sherri.smith@duke.edu) |
| Date or version (if downloaded, provide | Date of data pull (locked data): 10/17/2024 |
| date) | |
| Data transfer method and date | Direct data extraction from REDCap |
| Where dataset is stored | REDCap |
| | Extracted data and analytic datasets will be stored in |
| | a secure drive on the CRU folder. Path name: |
| | \\duhs-vclin- |
| | nc1\dusom_biostats_fs\Data\BiostatsCore\CRU\Head |
| | and Neck\Smith\PCORI_Pro00106077\Data pulls |

Notes: Additional variable details for all variables can be found in the "PCORI Variable Details" Excel file. Scoring details for APHAB can be found in "PCORI Scoring 20240923".

Description:

# 3 Outcomes, Exposures, and Additional Variables of Interest

### 3.1 Primary Outcome(s)

| Outcome | Description | Variables and Source | Specifications |
|---|---|---|---|
| APHAB Change<br>Score | Difference in aided APHAB scores at month 3 and unaided scores at baseline | aphab_change | Scale score – will need to calculate global communication scores at baseline (unaided) and 3 months (aided), subtract (3 months – baseline) A lower score on APHAB is better. |

| Rescore variables and multiply by 100 |
|---|
| <ul> <li>1 = 0.99</li> <li>2 = 0.87</li> <li>3 = 0.75</li> </ul> |
| <ul> <li>3 = 0.75</li> <li>4 = 0.50</li> <li>5 = 0.25</li> </ul> |
| <ul> <li>6 = 0.12</li> <li>7 = 0.01</li> </ul> |
| Reverse score questions 1, 9, 11, 16, 19, 21 |
| Global score: mean of variables in the EC, BN, RV subscale scores (excludes questions 3, 8, 13, 17, 20, 22) |
| Note: APHAB has 4 subscales and a global communication scale. The study is powered based on the benefit score on the global communication scale (August 2019 draft – APHAB SD of 25 with different levels of Cohen's |
| D). |

# 3.2 Secondary Outcome(s)

| Outcome | Description | Variables and Source | Specifications |
|---|---|---|---|
| APHAB change<br>score – binary, 3<br>months | Responders vs<br>non-<br>responders<br>for primary<br>APHAB<br>outcome | Decrease of 25 units: use aphab_change_responder Decrease of 15 units: use aphab_change_responder15 | Patients with a decrease of at least 25 units (or 15 units for the sensitivity analysis) on the APHAB scale at month 3 will be considered "responders." Patients not returning or who do not have a score at 3 months will be considered "non-responders." Patients with a baseline score < 25 (or < 15) are ineligible (missing). Binary (25 unit decrease): Missing if baseline score < 25 If aphab_change <=-25 |

| | | | <ul> <li>0 else</li> <li>Binary (15 unit decrease);</li> <li>Missing if baseline score &lt;15</li> <li>1 if aphab_change &lt;=-15</li> <li>0 else</li> </ul> |
|---|---|---|---|
| APHAB – 4 subscales | EC, BN, RV, AV scales at both baseline and 3 months, as well as change scores | Baseline variables: aphab_ec_base aphab_bn_base aphab_rv_base aphab_av_base 3-month variables: aphab_ec_3m aphab_bn_3m aphab_rv_3m Change scores: aphab_ec_change aphab_bn_change aphab_av_change aphab_av_change | Rescore variables and multiply by 100 1 = 0.99 2 = 0.87 3 = 0.75 4 = 0.50 5 = 0.25 6 = 0.12 7 = 0.01 Reverse score questions 1, 9, 11, 16, 19, 21 EC: mean of questions 4, 10, 12, 14, 15, 23 BN: mean of questions 1, 6, 7, 16, 19, 24 RV: mean of questions 2, 5, 9, 11, 18, 21 AV: mean of questions 3, 8, 13, 17, 20, 22 |

# 3.3 Additional Variables of Interest

| Variable | Description | Variables and Source | Specifications |
|---|---|---|---|
| Randomization assignment | Hearing aid assignment | assign | Binary 1: unilateral 2: bilateral |
| Clinical site | Which site -<br>Duke or<br>Vanderbilt? | which_site Character version: which_site_ch | Binary<br>1: Vanderbilt<br>2: Duke |
| Gender | | gender Character version: gender_ch | Categorical <ul><li>1: male</li><li>2: female</li><li>3: other</li><li>99: declined</li></ul> |
| Age | Age at baseline (years) | age_base | Continuous |

| | | Baseline visit is | Years from baseline_date |
|---|---|---|---|
| | | baseline_date | to dob |
| | | | Baseline visit is defined |
| | | | as aphab_base_date if |
| | | | non-missing, otherwise |
| | | | use date_moca |
| Race | | race | Categorical |
| | | | • 1: African |
| | | Character version: race_ch | American/Black |
| | | | <ul><li>2: White/Caucasian</li><li>3: Asian</li></ul> |
| | | | <ul><li>3: Asian</li><li>4: Native</li></ul> |
| | | | American/Alaska |
| | | | Native |
| | | | • 5: Native |
| | | | Hawaiian/Pacific |
| | | | Islander |
| | | | 6: More than one race |
| | | | • 99: Declined |
| | | | If cell counts are less |
| | | | than 10 for a given |
| | | | category, we may not |
| | | | report the exact cell count. |
| | | | count. |
| | | | NIH racial categories: |
| | | | -American Indian/Alaska |
| | | | Native |
| | | | -Asian or Asian American |
| | | | -Black or African |
| | | | American |
| | | | -Native Hawaiian/Pacific |
| | | | Islander |
| Ethnicity | | ethnicity | -White<br>Categorical |
| | | , | • 1: Hispanic or Latino |
| | | Character version: | 2: Not Hispanic or |
| | | ethnicity_ch | Latino |
| | | | 999: Declined |
| | | | If cell counts are less |
| | | | than 10 for a given |
| | | | category, we may not |
| | | | report the exact cell |
| Income | Personal | income | count. Categorical |
| income | Income Last | meonic | • 0: \$0 |
| | Year | Character version: | • 1: \$1 to \$9999 |
| | | income ch | • 2: \$10,000 to \$24,999 |
| | | _ | • 3: \$25,000 to \$49,999 |
| | | | • 4: \$50,000 to \$74,999 |

| Hearing Aid | | benefits | <ul> <li>5: \$75,000 to \$99,999</li> <li>6: \$100,000 to<br/>\$149,999</li> <li>7: \$150,000 or greater</li> <li>999: Prefer not to<br/>answer</li> <li>We will also simplify this<br/>to below median/above<br/>median/prefer not to<br/>answer for heterogeneity<br/>of treatment effects</li> <li>Categorical</li> </ul> |
|---|---|---|---|
| Health Insurance<br>Benefits | | Character version: benefits_ch | <ul><li>0: No</li><li>1: Yes</li><li>998: Not Sure</li></ul> |
| Marital Status | | marital Character version: marital_ch | Categorical 1: married 2: widowed 3: divorced 4: separated 5: never married 999: prefer not to answer |
| Living arrangements | | living Character version: living_ch | Categorical 1: alone 2: with spouse 3: with spouse and others 888: other 999: prefer not to answer |
| Education | | education Character version: education_ch | Categorical 1: less than high school 2: high school 3: some college 4: 4-year degree 5: graduate degree 888: other 999: prefer not to answer |
| Baseline Date<br>Quarter | | baseline_quarter | Categorical Put baseline date into quarters |
| Cognition<br>(Screened via<br>MoCA) | Adjusted<br>MoCA score | total_moca | Continuous, 0-30 moca31 is a modifier for high school education |

| | | | If moca31=0, then total moca score is the sum of moca1 through moca30 If moca31=1, then total moca score is the minimum of 30 and the sum of moca1 through |
|---|---|---|---|
| Audiogram Data | Frequencies: 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000, 8000, 12000 Create a "complete" audiogram using screening and baseline data | Right ear (numeric): audio_r_250_unaided audio_r_500_unaided audio_r_1000_unaided audio_r_1500_unaided audio_r_2000_unaided audio_r_3000_unaided audio_r_4000_unaided audio_r_6000_unaided audio_r_12000_unaided audio_r_12000_unaided audio_r_12000_unaided audio_l_500_unaided audio_l_1500_unaided audio_l_1500_unaided audio_l_1500_unaided audio_l_1500_unaided audio_l_16000_unaided audio_l_9000_unaided audio_l_9000_unaided audio_l_1000_unaided audio_r_500_unaided_nr audio_r_1500_unaided_nr audio_r_1000_unaided_nr | moca 31 Will create a "complete" audiogram by combining baseline and screening visit audiograms — baseline visit takes priority over screening visit. Variables are originally stored as character — can have responses like "NA", "NR", "DNT". Convert to numeric. If we have any responses like this, set to missing. If "NR" — create a flag for each frequency and each ear to be 1 (0 else) |

| | | audio_l_750_unaided_nr<br>audio_l_1000_unaided_nr<br>audio_l_1500_unaided_nr<br>audio_l_2000_unaided_nr<br>audio_l_3000_unaided_nr<br>audio_l_4000_unaided_nr<br>audio_l_6000_unaided_nr<br>audio_l_8000_unaided_nr<br>audio_l_12000_unaided_nr | |
|---|---|---|---|
| Degree of Hearing Loss – Pure Tone Average | PTA in better<br>ear | Right ear: pta_right Left ear: pta_left Better ear: pta_better | We will use the pure tone average in the better ear. Take the average at frequencies 500, 1000, 2000, 4000 in both ears. The lower average is the better ear. |
| Hearing loss classification | | hearing_loss_class | <ul> <li>Mild: pta_better &lt;= 40</li> <li>Moderate pta_better &gt; 40</li> </ul> |

# 4 Statistical Analysis Plan

Analysis: To be completed by December 31, 2024

### 4.1 Demographic and Clinical Characteristics ("Table 1")

Analysis: This will be descriptive. As appropriate, we will present the mean with standard deviation (SD), median with interquartile range (IQR), and ranges (min and max), or frequency with percentage (see Table 1). Categorical variables may be collapsed into fewer categories. If cell counts are less than 10 for variables that could identify patients (e.g., race, ethnicity), we may not report the exact cell count. We may consider stratifying this table by clinical site as well.

| Table 1: Patient Characteristics at Baseline | | | |
|---|---|---|---|
| | Unilateral<br>(N=XXX) | Bilateral<br>(N=XXX) | Total<br>(N=XXX) |
| Clinical Site | | | |
| Duke | XXX (%) | XXX (%) | XXX (%) |
| Vanderbilt | XXX (%) | XXX (%) | XXX (%) |
| Gender | | | |
| Female | XXX (%) | XXX (%) | XXX (%) |
| Male | XXX (%) | XXX (%) | XXX (%) |
| Other | XXX (%) | XXX (%) | XXX (%) |
| Age at Baseline Visit | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |

| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
|---------------------------------------|-----------|-----------|-----------|
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX , XXX | XXX , XXX | XXX , XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| Race | 7000 7000 | 7000 7000 | 7000 7000 |
| American Indian/Alaska Native | XXX (%) | XXX (%) | XXX (%) |
| Asian | XXX (%) | XXX (%) | XXX (%) |
| Black or African American | XXX (%) | XXX (%) | XXX (%) |
| White | XXX (%) | XXX (%) | XXX (%) |
| More than one race | XXX (%) | XXX (%) | XXX (%) |
| Native Hawaiian/Pacific Islander | XXX (%) | XXX (%) | XXX (%) |
| Declined | XXX (%) | XXX (%) | XXX (%) |
| Ethnicity | , | , | ( ) |
| Hispanic or Latino | XXX (%) | XXX (%) | XXX (%) |
| Not Hispanic or Latino | XXX (%) | XXX (%) | XXX (%) |
| Declined | XXX (%) | XXX (%) | XXX (%) |
| Personal Income Last Year | , , | , , | , , |
| \$0 | XXX (%) | XXX (%) | XXX (%) |
| \$1 to \$9999 | XXX (%) | XXX (%) | XXX (%) |
| \$10,000 to \$24,999 | XXX (%) | XXX (%) | XXX (%) |
| \$25,000 to \$49,999 | XXX (%) | XXX (%) | XXX (%) |
| \$50,000 to \$74,999 | XXX (%) | XXX (%) | XXX (%) |
| \$75,000 to \$99,999 | XXX (%) | XXX (%) | XXX (%) |
| \$100,000 to \$149,999 | XXX (%) | XXX (%) | XXX (%) |
| \$150,000 or greater | XXX (%) | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) | XXX (%) |
| Personal Income Last Year | | | |
| (Categorical) | | | |
| Below Median | XXX (%) | XXX (%) | XXX (%) |
| Above Median | XXX (%) | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) | XXX (%) |
| Hearing Aid Health Insurance Benefits | | | |
| No | XXX (%) | XXX (%) | XXX (%) |
| Yes | XXX (%) | XXX (%) | XXX (%) |
| Not sure | XXX (%) | XXX (%) | XXX (%) |
| Marital Status | | | |
| Married | XXX (%) | XXX (%) | XXX (%) |
| Widowed | XXX (%) | XXX (%) | XXX (%) |
| Divorced | XXX (%) | XXX (%) | XXX (%) |
| Separated | XXX (%) | XXX (%) | XXX (%) |
| Never married | XXX (%) | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) | XXX (%) |
| Living Arrangements | | | |
| Alone | XXX (%) | XXX (%) | XXX (%) |
| With spouse | XXX (%) | XXX (%) | XXX (%) |

| With spouse and others | XXX (%) | XXX (%) | XXX (%) |
|------------------------------------------|-----------|-----------|-----------|
| Other | XXX (%) | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) | XXX (%) |
| Education | | | |
| Less than high school | XXX (%) | XXX (%) | XXX (%) |
| High school | XXX (%) | XXX (%) | XXX (%) |
| Some college | XXX (%) | XXX (%) | XXX (%) |
| 4-year degree | XXX (%) | XXX (%) | XXX (%) |
| Graduate degree | XXX (%) | XXX (%) | XXX (%) |
| Other | XXX (%) | XXX (%) | XXX (%) |
| Quarter of Baseline Visit | | | |
| 2021 Q2 | XXX (%) | XXX (%) | XXX (%) |
| 2021 Q3 | XXX (%) | XXX (%) | XXX (%) |
| 2021 Q4 | XXX (%) | XXX (%) | XXX (%) |
| | XXX (%) | XXX (%) | XXX (%) |
| Total MoCA Score | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| Pure Tone Average in Better Ear** | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| Hearing Loss Classification in Better Ea | r | | |
| Mild | XXX (%) | XXX (%) | XXX (%) |
| Moderate | XXX (%) | XXX (%) | XXX (%) |

We will create a table for clinical characteristics (Supplemental Table 1) which will be given to Sherri Smith in order to create an audiogram that follows the standards of the field.

<sup>\*\*</sup>Average value for frequencies of 500, 1000, 2000, 4000 Hz

| | Unilateral | Bilateral | Total |
|--------------------|------------|-----------|-----------|
| | (N=XXX) | (N=XXX) | (N=XXX) |
| Right Ear: 250 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 500 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 750 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 1000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 1500 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 2000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 3000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 4000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 6000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Right Ear: 8000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| | XXX | XXX | XXX |

| N | XXX | XXX | XXX |
|--------------------|-----------|-----------|-----------|
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 250 Hz | 7000 | 7000 | 7000 |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 500 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 750 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 1000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 1500 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 2000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 3000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 4000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 6000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 8000 Hz | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| Left Ear: 12000 Hz | | | |

| N | XXX | XXX | XXX |
|-------------------------------|-----------|-----------|-----------|
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| NR Values | XXX | XXX | XXX |
| (report generated on XXXXXXX) | | | |

### 4.2 Describe APHAB Global Score Distributions and Responder Status

We will describe the distribution of APHAB global score at baseline (unaided) and 3 months (aided), along with the change score and responder status (both definitions) by hearing aid assignment in Table 2.

| | Unilateral | Bilateral | Total |
|-------------------------------|------------|-----------|-----------|
| | (N=XXX) | (N=XXX) | (N=XXX) |
| APHAB Global Score (Baseline) | | | • |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB Global Score (3 Months) | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB Change Score | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB Responder (25 Units)* | | | |
| No | XXX (%) | XXX (%) | XXX (%) |
| Yes | XXX (%) | XXX (%) | XXX (%) |
| Ineligible to Drop 25 Units | XXX | XXX | XXX |
| APHAB Responder (15 Units)* | | | |
| No | XXX (%) | XXX (%) | XXX (%) |
| Yes | XXX (%) | XXX (%) | XXX (%) |
| Ineligible to Drop 15 Units | XXX | XXX | XXX |

### 4.3 Primary aim: compare APHAB scores between the two arms

Compare the APHAB change scores between the two arms (bilateral hearing aid and unilateral hearing aid) at the end of month 3 vs baseline.

Analysis: This will be done for all randomized patients who have both baseline and 3 month scores (a "completers" analysis). The primary analysis will be performed by linear regression and include randomized assignment and clinical site as covariates.

APHAB change score = 
$$\beta_0 + \beta_1 * treatment + \beta_2 * site$$

| Table 3: Linear Regression Beta Estimat<br>Outcome Modelled: APHAB Cha | | | |
|---|---|---|---|
| Covariate | Beta | 95% C.I. | P-Value* |
| Hearing Aid Assignment (Reference: | | | |
| Bilateral) | | | |
| Unilateral | XXX | (XXX, XXX) | XXX |
| Clinical Site (Reference: Duke) | | | |
| Vanderbilt | XXX | (XXX, XXX) | XXX |
| *Using XXX statistic | | | |

### 4.4 Heterogeneity of Treatment Effects Analysis for APHAB scores

Compare APHAB change scores between the two arms at the end of month 3 vs baseline while adjusting for interaction terms between treatment and each variable of interest.

Analysis: This will be done for all randomized patients who have both baseline and 3 month scores ("completers"). The primary analysis will be performed by linear regression and include randomized assignment, clinical site, a given variable of interest (denoted by S), and interactions between treatment and the variable of interest, with separate models fit for each variable of interest. The two variables of interest that decided to investigate are income group (simplified version – below median, above median, prefer not to answer) and hearing loss classification (mild, moderate). Interactions will be tested at the 0.15 level. If the overall test for the interaction is significant, forest plots will be constructed to examine the heterogeneity of treatment effect and formal treatment by factor interaction terms tested in the models. The general model structure is:

APHAB change score = 
$$\beta_0 + \beta_1 * treatment + \beta_2 * site + \beta_S * S + \beta_{ST} * S * treatment$$

| Table 4: Linear Regression Beta Estimates for Variable S Model Outcome Modelled: APHAB Change Score | | | |
|---|---|---|---|
| Covariate | Beta | 95% C.I. | P-Value* |
| Hearing Aid Assignment (Reference: | | | |
| Bilateral) | | | |
| Unilateral | XXX | (XXX, XXX) | XXX |
| Clinical Site (Reference: Duke) | | | |
| Vanderbilt | XXX | (XXX, XXX) | XXX |
| Variable S | XXX | (XXX, XXX) | XXX |
| HA Assignment*Variable S | XXX | (XXX, XXX) | XXX |

#### 4.5 Sensitivity analyses for APHAB scores

If more than 5% of randomized patients have missing APHAB scores at 3 months, we will use multiple imputation in an intent to treat sensitivity analysis.

Analysis 1: An imputation model via linear regression will be developed based on available data and will include initial APHAB scores, treatment, baseline characteristics, and possible interactions of these variables with treatment. The specific variables of interest to include are: treatment, site, income group, and baseline APHAB. A total of 1000 datasets with imputations of APHAB score reduction will be generated using this model. Each dataset will be analyzed using linear regression models as described in section 4.3. The combined results will be reported and will take the variability of multiple imputations into account.

Analysis 2: The characteristics from the participants with completed data will be compared to those with missing APHAB data with the use of a "Table 1". We may also include treatment randomization in this table.

| | Missing APHAB | Not Missing APHAB | |
|---|---|---|---|
| | (N=XXX) | (N=XXX) | Total (N=XXX) |
| Assignment | | | |
| Unilateral | XXX (%) | XXX (%) | XXX (%) |
| Bilateral | XXX (%) | XXX (%) | XXX (%) |
| Clinical Site | | | |
| Duke | XXX (%) | XXX (%) | XXX (%) |
| Vanderbilt | XXX (%) | XXX (%) | XXX (%) |
| Gender | | | |
| Female | XXX (%) | XXX (%) | XXX (%) |
| Male | XXX (%) | XXX (%) | XXX (%) |
| Other | XXX (%) | XXX (%) | XXX (%) |
| Age at Baseline Visit | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| Race | | | |
| American Indian/Alaska Native | XXX (%) | XXX (%) | XXX (%) |
| Asian | XXX (%) | XXX (%) | XXX (%) |
| Black or African American | XXX (%) | XXX (%) | XXX (%) |
| White | XXX (%) | XXX (%) | XXX (%) |
| More than one race | XXX (%) | XXX (%) | XXX (%) |
| Native Hawaiian/Pacific Islander | XXX (%) | XXX (%) | XXX (%) |
| Declined | XXX (%) | XXX (%) | XXX (%) |

| Historia au Latina | VVV (0/) | VVV (0/) | VVV (0/) |
|---|---|---|---|
| Hispanic or Latino Not Hispanic or Latino | XXX (%)<br>XXX (%) | XXX (%)<br>XXX (%) | XXX (%) |
| Declined | XXX (%) | XXX (%) | XXX (%)<br>XXX (%) |
| Personal Income Last Year | AAA (70) | AAA (70) | AAA (70) |
| \$0 | XXX (%) | XXX (%) | XXX (%) |
| \$1 to \$9999 | XXX (%) | XXX (%) | XXX (%) |
| \$10,000 to \$24,999 | XXX (%) | XXX (%) | XXX (%) |
| \$25,000 to \$49,999 | XXX (%) | XXX (%) | XXX (%) |
| \$50,000 to \$74,999 | XXX (%) | XXX (%) | XXX (%) |
| \$75,000 to \$99,999 | XXX (%) | XXX (%) | XXX (%) |
| \$100,000 to \$149,999 | XXX (%) | XXX (%) | XXX (%) |
| \$150,000 or greater | XXX (%) | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) | XXX (%) |
| Personal Income Last Year | XXX (70) | XXX (70) | XXX (70) |
| (Categorical) | | | |
| Below Median | XXX (%) | XXX (%) | XXX (%) |
| Above Median | XXX (%) | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) | XXX (%) |
| Hearing Aid Health Insurance | ( , | (* ) | ( , |
| Benefits | | | |
| No | XXX (%) | XXX (%) | XXX (%) |
| Yes | XXX (%) | XXX (%) | XXX (%) |
| Not sure | XXX (%) | XXX (%) | XXX (%) |
| Marital Status | | | |
| Married | XXX (%) | XXX (%) | XXX (%) |
| Widowed | XXX (%) | XXX (%) | XXX (%) |
| Divorced | XXX (%) | XXX (%) | XXX (%) |
| Separated | XXX (%) | XXX (%) | XXX (%) |
| Never married | XXX (%) | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) | XXX (%) |
| Living Arrangements | | | |
| Alone | XXX (%) | XXX (%) | XXX (%) |
| With spouse | XXX (%) | XXX (%) | XXX (%) |
| With spouse and others | XXX (%) | XXX (%) | XXX (%) |
| Other | XXX (%) | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) | XXX (%) |
| Education | | | |
| Less than high school | XXX (%) | XXX (%) | XXX (%) |
| High school | XXX (%) | XXX (%) | XXX (%) |
| Some college | XXX (%) | XXX (%) | XXX (%) |
| 4-year degree | XXX (%) | XXX (%) | XXX (%) |
| Graduate degree | XXX (%) | XXX (%) | XXX (%) |
| Other | XXX (%) | XXX (%) | XXX (%) |
| Quarter of Baseline Visit | | | |
| 2021 Q2 | XXX (%) | XXX (%) | XXX (%) |

| 2021 Q3 | XXX (%) | XXX (%) | XXX (%) |
|-----------------------------|-----------|-----------|-----------|
| m | XXX (%) | XXX (%) | XXX (%) |
| Total MoCA Score | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| Pure Tone Average in Better | Ear | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| Hearing Loss Classification | | | |
| Mild | XXX (%) | XXX (%) | XXX (%) |
| Moderate | XXX (%) | XXX (%) | XXX (%) |
| (report generated on XXXXXX | X) | | |

Analysis 3: We will report the rate of dropout in each of the two groups and look at the potential imbalances in dropouts between randomized interventions. We will report clinically meaningful differences. Given the size of the study, the ability to detect MNAR is small.

#### 4.6 Analyze APHAB binary response at 3 months

Patients with a decrease of at least 25 units on the APHAB scale at month 3 compared to baseline unaided APHAB will be defined as "responders." Patients who do not meet this criterion of 25 units, do not return, or do not have a score at month 3 will be defined as "non-responders." If there are any patients with unaided APHAB scores of less than 25, these patients will be excluded as they are not eligible to drop 25 units.

**Analysis 1:** This will be done for all randomized patients who are eligible, including those missing APHAB change scores. This analysis will be performed by logistic regression and include randomized assignment and clinical site as covariates.

Binary APHAB change  $score = \beta_0 + \beta_1 * treatment + \beta_2 * site$ 

| Table 6: Logistic Regression OR Estimates Outcome Modelled: Binary APHAB Change Score Response (25 Unit) | | | |
|---|---|---|---|
| Covariate | OR | 95% C.I. | P-Value* |
| Hearing Aid Assignment (Reference: | | | |
| Bilateral) | | | |
| Unilateral | XXX | (XXX, XXX) | XXX |
| Clinical Site (Reference: Duke) | | | |
| Vanderbilt | XXX | (XXX, XXX) | XXX |

\*Using XXX statistic

Analysis 2 (heterogeneity of treatment effects): This analysis will be performed by logistic regression and include randomized assignment, clinical site, a given variable of interest (denoted by S), and interactions between treatment and the variable of interest, with separate models fit for each variable of interest. The two variables of interest that decided to investigate are income group (simplified version – below median, above median, prefer not to answer) and hearing loss classification (mild, moderate). Interactions will be tested at the 0.15 level. If the overall test for the interaction is significant, forest plots will be constructed to examine the heterogeneity of treatment effect and formal treatment by factor interaction terms tested in the models. The general model structure is:

Binary APHAB change score =  $\beta_0 + \beta_1 * treatment + \beta_2 * site + \beta_S * S + \beta_{ST} * S * treatment$ 

We will report the joint test p-value for the interaction term. If significant, we will report odds ratios and 95% confidence intervals.

| Covariate | OR | 95% C.I. | P-Value* |
|------------------------------------|-----|------------|----------|
| Hearing Aid Assignment (Reference: | | | |
| Bilateral) | | | |
| Unilateral | XXX | (XXX, XXX) | XXX |
| Clinical Site (Reference: Duke) | | | |
| Vanderbilt | XXX | (XXX, XXX) | XXX |
| Variable S | XXX | (XXX, XXX) | XXX |
| HA Assignment*Variable S | XXX | (XXX, XXX) | XXX |

Analyses 3-4: repeat analyses 1-2 of this section, but define responders as having a decrease of at least 15 units.

Binary APHAB change score =  $\beta_0 + \beta_1 * treatment + \beta_2 * site$ 

| Outcome Modelled: Binary APH | AB Change Scor | e (15 Unit) | |
|------------------------------------|----------------|-------------|----------|
| Covariate | OR | 95% C.I. | P-Value* |
| Hearing Aid Assignment (Reference: | | | |
| Bilateral) | | | |
| Unilateral | XXX | (XXX, XXX) | XXX |
| Clinical Site (Reference: Duke) | | | |
| Vanderbilt | XXX | (XXX, XXX) | XXX |

Binary APHAB change score =  $\beta_0 + \beta_1 * treatment + \beta_2 * site + \beta_S * S + \beta_{ST} * S * treatment$ 

| Table 9 Logistic Regression | OR Estimates for Variable S | Model | |
|---|---|---|---|
| Outcome Modelled | l: Binary APHAB Change Score | e (15 Unit) | |
| Covariate | Beta | 95% C.I. | P-Value* |

| Hearing Aid Assignment (Reference: | | | |
|------------------------------------|-----|------------|-----|
| Bilateral) | | | |
| Unilateral | XXX | (XXX, XXX) | XXX |
| Clinical Site (Reference: Duke) | | | |
| Vanderbilt | XXX | (XXX, XXX) | XXX |
| Variable S | XXX | (XXX, XXX) | XXX |
| HA Assignment*Variable S | XXX | (XXX, XXX) | XXX |
| *Using XXX statistic | | 301 | |

### 4.7 Describe APHAB Subscales

We will describe the distribution of the 4 APHAB subscales (EC, BN, RV, AV) at baseline (unaided) and 3 months (aided) by hearing aid assignment, along with the change scores graphically and in a Table (Table 10).

| | Unilateral | Bilateral | Total |
|--------------------------------|------------|-----------|-----------|
| | (N=XXX) | (N=XXX) | (N=XXX) |
| APHAB EC Subscale (Baseline) | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB EC Subscale (3 Months) | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB EC Subscale Change Score | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB BN Subscale (Baseline) | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |

| APHAB BN Subscale (3 Months) | | | |
|--------------------------------|-----------|-----------|-----------|
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB BN Subscale Change Score | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB RV Subscale (Baseline) | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB RV Subscale (3 Months) | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB RV Subscale Change Score | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB AV Subscale (Baseline) | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB AV Subscale (3 Months) | | | |
| N | XXX | XXX | XXX |

| Missing | XXX | XXX | XXX |
|--------------------------------|-----------|-----------|-----------|
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| APHAB AV Subscale Change Score | | | |
| N | XXX | XXX | XXX |
| Missing | XXX | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX | XXX - XXX |
| (report generated on XXXXXXX) | | | |

### 4.8 Initially planned analyses that we will not do

We had initially planned to conduct adjusted analyses for the outcomes of global change score and both responder definitions. After reviewing cell counts of demographics at baseline and discussion, we decided that there are no variables of interest to include in an adjusted model.

# Statistical Analysis Plan (SAP) – Secondary (3-Month) Outcomes and Descriptives

**Project:** Evaluation of Unilateral vs Bilateral Hearing Aids for the Treatment of Age-related Hearing

Loss

IRB Number: Pro00106077

Investigator(s): Sherri Smith, AuD, PhD

Biostatistician(s): Kayla Kilpatrick, PhD, Sarah Peskoe, PhD, Frank Rockhold, PhD

**Original Creation Date: 12.15.2021** 

Version Date: 09.30.2024

| Investigator Agreement | reflect the wo changes or ad findings without All biostatistic review the ful included as conthe analyses. If substantial approject change Publications reduced CTSA and submitted to It have reviewed documented. Acknowledged by | analyses included in an abstract or manuscript should ork of the biostatistician(s) listed on this SAP. No ditional analyses should be made to the results or out discussing with the project biostatistician(s). Scians on this SAP should be given sufficient time to I presentation, abstract, manuscript, or grant and be reauthors on any abstract or manuscript resulting from additional analysis is necessary or the aims of the e, a new SAP will need to be developed. Esulting from this SAP are supported in part by the d must cite grant number UL1TR002553 and be PubMed Central. End the SAP and understand that any changes must be expected or the same of t |
|---|---|---|
| Activity Log | 05.31.2024 Adde<br>07.11.2024 Reso<br>20240531 and O<br>07.25.2024 Mov | secondary outcomes SAP into multiple SAPs ed additional variables blved some questions about variables (see SAP dated everview of All Planned Analysis dated 20240620) ed GHABP from the GHABP/EMA SAP to this SAP ated variable names, resolved comments from previous 0725) |
| Acronyms | APHAB<br>EMA<br>GHABP<br>IOI-HA<br>SADL<br>SSQ<br>HHIE | Abbreviated Profile of Hearing Aid Benefit Ecological Momentary Assessment Glasgow Hearing Aid Benefit Profile International Outcomes Inventory for Hearing Aids Satisfaction with Amplification in Daily Life Speech Spatial Qualities Hearing Handicap Inventory for Elderly |

## 1 Study Overview

Background/Introduction: The overall goal of the project is to determine the benefit of unilateral or bilateral hearing aid fittings in adults with mild-to-moderate age-related hearing loss. This will address the lack of high-quality evidence supporting bilateral hearing aids over unilateral hearing aids. This project will use a randomized controlled trial with two treatment arms: a bilateral hearing aid fitting group and a unilateral hearing aid fitting group.

#### 1.1 Aims for Secondary Outcomes

- Compare all outcomes between the two arms (bilateral hearing aid and unilateral hearing aid) at 3 months. The primary hypothesis is that bilateral hearing aids are superior to the unilateral hearing aids with respect to the overall patient-reported benefit.
- Descriptive tables for additional clinical variables at baseline and 3-months by assigned treatment
- Plots of hearing aid fit by assigned treatment

# 2 Study Population

#### 2.1 Inclusion Criteria

- 50+ years of age
- Mild to moderate, symmetrical SNHL (symmetrical: < 20 dB between ears on average from 500-4000 Hz)
- Open-mindedness to unilateral or bilateral amplification
- No prior hearing aid experience
- Adequate literacy to complete questionnaires
- Willing to purchase study-specific hearing aid(s)

#### 2.2 Exclusion Criteria

- Concerns for middle ear pathology
- Concerns for retrocochlear pathology
- Severe tinnitus as the reason for seeking amplification
- Co-morbid condition that would interfere with study (e.g., dementia, blindness, neurologic pathology)
- History of fluctuating hearing loss

### 2.3 Data Acquisition

Fill in all relevant information:

| Study design | Randomized controlled trial with 2 arms (bilateral hearing aid, unilateral hearing aid) |
|---|---|
| | Note: Randomization was stratified by clinical site. |
| Data source/how the data were collected | Screening information pulled from EHR data |
| butu source/now the data were concered | Baseline surveys captured via in-person interview and recorded in REDCap |
| Contact information for team member | All data access is through |
| responsible for data | . Questions on data validity |
| collection/acquisition | will go to PI: Sherri Smith (Sherri.smith@duke.edu) |
| Date or version (if downloaded, provide | 10.17.2024 |
| date) | |
| Data transfer method and date | Direct data extraction from REDCap |
| Where dataset is stored | REDCap |

Extracted data and analytic datasets are stored on a secure drive in the CRU folder: \\duhs-vclin-nc1\dusom biostats fs\Data\BiostatsCore\CRU\Head and Neck\Smith\PCORI Pro00106077\Data pulls

Notes: Additional variable details for all variables can be found in the "PCORI Variable Details" Excel file. Scoring details can be found in "PCORI Scoring 20240923".

#### For GHABP:

6 total scenarios, 4 standard, 2 user-nominated. Standard scenarios:

- 1. LISTENING TO THE TELEVISION WITH OTHER FAMILY OR FRIENDS WHEN THE VOLUME IS ADJUSTED TO SUIT OTHER PEOPLE
- 2. HAVING A CONVERSATION WITH ONE OTHER PERSON WHEN THERE IS NO BACKGROUND NOISE
- 3. CARRYING ON A CONVERSATION IN A BUSY STREET OR SHOP
- 4. HAVING A CONVERSATION WITH SEVERAL PEOPLE IN A GROUP

### **Unaided questions:**

- 1. Does this situation happen in your life?
- 2. How much difficulty do you have in this situation?
- 3. How much does any difficulty in this situation worry, annoy or upset you?

### Aided/EMA questions:

- 1. Did this situation happen in the past few weeks? (GHABP aided) OR Did this situation happen in the last three hours? (EMA)
- 2. In this situation, with your hearing aid, how much does any difficulty in this situation worry, annoy or upset you? NOTE: this question is non-standard for the aided GHABP. We will report on this in a descriptive table but will not include in analyses.
- 3. In this situation, what proportion of the time do you wear your hearing aid?
- 4. In this situation, how much does your hearing aid help you?
- 5. In this situation, with your hearing aid, how much difficulty do you now have?
- 6. For this situation, how satisfied are you with your hearing aid?

### Description:

# 3 Outcomes, Exposures, and Additional Variables of Interest

### 3.1 Outcome(s)

| Outcome | Description | Variables and Source | Specifications |
|---|---|---|---|
| IOI-HA | Note: this is<br>measured<br>only at 3 and<br>6 months | Total score: ioiha_total_3m | Total score: sum responses to questions 1-7 (should be on a range between 1-5). |
| | | | Item 8 is self-perceived hearing difficulty used for normative purposes |

| | | | (currently not used as part of total score) This is initially coded as 0 to 4 in REDCap — changed to 1-5 Currently, we're treating IOI-HA total score as continuous, but this may need to be treated as ordinal. |
|---|---|---|---|
| | | | Higher scores are better |
| SADL | Note: this is measured only at 3 and 6 months. Note: the "sister" questionnaire at baseline is ECHO | Positive effect subscale: sadl_positive_effect_3m Service cost subscale: sadl_service_cost_3m Negative features subscale: sadl_negative_features_3m Personal image subscale: sadl_personal_image_3m | Questions 1 – 15 are used. This is scored from 1-7 (or reversed for questions 2, 4, 7, 13). There are 4 subscales: Positive Effect, Service & Cost, Negative Features, Personal Image. For each subscale, the average score is calculated. For the global score, this is the mean of the scores for all items (excluding questions 11 and 14 if applicable). Higher scores are better (higher satisfaction). See PCORI Scoring file for more details |
| SSQ | Note: this is measured at baseline, 3 months, and 6 months. | Change score: ssq_change Baseline: Overall score: ssq_overall_base Speech/hearing subscale: ssq_speech_hearing_base Spatial/hearing subscale: ssq_spatial_hearing_base | 3 subscales: Speech is questions 1 – 14 (corresponds to the "pt1" variables). Spatial is 17 questions (corresponds to the "pt2" variables). Qualities is 18 questions (correspond to the "pt3" variables). |

| 3-Months: Overall score: ssq_overall_3m Speech/hearing subscale: ssq_speech_hearing_3m Spatial/hearing subscale: ssq_spatial_hearing_3m Qualities of hearing_3m Qualities_of_hearing_3m Sq_qualities_of_hearing_3m We will also create a change score as the difference in the overall score between 3 months and baseline (3 months – baseline) Higher scores are better | i | | Qualities of hearing subscale: | Overall score: mean of |
|---|---|---|---|---|
| Overall score: ssq_overall_3m Speech/hearing subscale: ssq_speech_hearing_3m Spatial/hearing subscale: ssq_spatial_hearing_3m Qualities of hearing subscale: ssq_qualities_of_hearing_3m Qualities_of_hearing_3m We will also create a change score as the difference in the overall score between 3 months and baseline (3 months – baseline) Higher scores are better | | | ssq_qualities_of_hearing_base | the items. |
| Overall score: ssq_overall_3m Speech/hearing subscale: ssq_speech_hearing_3m Spatial/hearing subscale: ssq_spatial_hearing_3m Qualities of hearing subscale: ssq_qualities_of_hearing_3m Qualities_of_hearing_3m We will also create a change score as the difference in the overall score between 3 months and baseline (3 months – baseline) Higher scores are better | | | 2-Months: | For instances where |
| speech/hearing subscale: ssq_speech_hearing_3m Spatial/hearing subscale: ssq_spatial_hearing_3m Qualities of hearing subscale: ssq_qualities_of_hearing_3m We will also create a change score as the difference in the overall score between 3 months and baseline (3 months – baseline) Higher scores are better | | | ' <del></del> | |
| ssq_speech_hearing_3m Spatial/hearing subscale: ssq_spatial_hearing_3m We will also create a change score as the difference in the overall score between 3 months and baseline (3 months – baseline) Higher scores are better | | | | • |
| Spatial/hearing subscale: ssq_spatial_hearing_3m We will also create a change score as the Qualities of hearing subscale: ssq_qualities_of_hearing_3m score between 3 months and baseline (3 months – baseline) Higher scores are better | | | Speech/hearing subscale: | set as NA. If a value |
| Spatial/hearing subscale: ssq_spatial_hearing_3m We will also create a change score as the difference in the overall ssq_qualities_of_hearing_3m score between 3 months and baseline (3 months – baseline) Higher scores are better | | | ssq_speech_hearing_3m | • |
| ssq_spatial_hearing_3m Ssq_spatial_hearing_3m Qualities of hearing subscale: ssq_qualities_of_hearing_3m score between 3 months and baseline (3 months – baseline) Higher scores are better | | | Castist the said and because | value. |
| Qualities of hearing subscale: ssq_qualities_of_hearing_3m score between 3 months and baseline (3 months – baseline) Higher scores are better | | | _ · | Wo will also create a |
| Qualities of hearing subscale: ssq_qualities_of_hearing_3m score between 3 months and baseline (3 months – baseline) Higher scores are better | | | ssq_spatiai_fleafflig_5fff | |
| ssq_qualities_of_hearing_3m score between 3 months and baseline (3 months – baseline) Higher scores are better | | | Qualities of hearing subscale: | difference in the overall |
| months – baseline) Higher scores are better | | | _ | score between 3 |
| Higher scores are better | | | | · · |
| | | | | months – baseline) |
| | | | | Higher scores are better |
| HHI-E Note: this is Change score: hhie_change Yes = 4 points, | HHI-E | Note: this is | Change score: hhie_change | _ |
| measured at Sometimes = 2 points, | | measured at | | Sometimes = 2 points, |
| baseline, 3 <u>Baseline</u> : and No = 0 points. | | • | · | and No = 0 points. |
| months, and 6 Total score: hhie_total_base | | - | Total score: hhie_total_base | Total cools coors – cors |
| months Situational subscale: Total scale score = sum of all 25 items | | months | Situational subscale: | |
| hhie situational base | | | | or all 23 feems |
| Situational subscale: | | | | Situational subscale: |
| Emotional subscale: questions 1, 3, 6, 8, 10, | | | Emotional subscale: | questions 1, 3, 6, 8, 10, |
| hhie_emotional_base 11 13, 15, 16, 19, 21, 23 | | | hhie_emotional_base | 11 13, 15, 16, 19, 21, 23 |
| 3-Months: Emotional subscale: | | | 3-Months: | Emotional subscale: |
| Total score: hhie_total_3m questions 2, 4, 5, 7, 9, | | | ' | |
| 12, 14, 17, 18, 20, 22, | | | | · · |
| Situational subscale: 24, 25 | | | Situational subscale: | 24, 25 |
| hhie_situational_3m | | | hhie_situational_3m | NA7 - 111 - 1 |
| We will also create a Emotional subscale: change score as the | | | Emotional subscalar | |
| hhie emotional 3m difference in the total | | | | • |
| scale score between 3 | | | | |
| months and baseline (3 | | | | months and baseline (3 |
| months – baseline) | | | | months – baseline) |
| Lower scores are hetter | | | | Lower scores are better |
| GHABP Aided Aided: 3 Question 2 average, 4 For questions 3-6 (IF | GHABP Aided | Aided: 3 | Question 2 average, 4 | |
| months standard scenarios: they answer yes to | | months | standard scenarios: | - |
| ghabp_q2_4block_3m question 1), doing this | | | ghabp_q2_4block_3m | |
| separately by question: | | | Ougstion 2 suggest 4 | |
| Question 3 average, 4 1. Subtract 1, standard scenarios: multiply by 25, | | | | · |
| ghabp_q3_4block_3m average answer | | | | • • • |
| to question across | | | | |

| | | Question 4 average, 4 | 4 standard |
|---|---|---|---|
| | | standard scenarios: | scenarios |
| | | ghabp_q4_4block_3m | Notorianoro current |
| | | | Note: ignore current question 2 for analyses |
| | | Question 5 average, 4 | as it is non-standard |
| | | standard scenarios: | but report on this in a |
| | | ghabp_q5_4block_3m | descriptive table |
| | | | descriptive table |
| | | Question 6 average, 4 | There are 6 scenarios (4 |
| | | standard scenarios: | standard, 2 user- |
| | | ghabp_q6_4block_3m | nominated) |
| | | | , |
| | | | Note that question 1 |
| | | | just asks if this scenario |
| | | | has happened – |
| | | | participants are only |
| | | | included in the |
| | | | averages if they answer |
| | | | "yes" |
| | | | Higher/lower seeres are |
| | | | Higher/lower scores are better depending on |
| | | | question |
| Speech and | Baseline | Baseline: | Continuous |
| Noise Test | (unaided) and | sin collocated base | Continuous |
| 110136 1636 | 3-months | sin right base | Change scores: 3m- |
| | (aided) | sin left base | baseline for each of |
| | (* * | | collocated, speech |
| | Speech and | 3-Months: | left/noise right, noise |
| | noise 0 | sin_collocated_3m | left/speech right |
| | degrees | sin_right_3m | |
| | (collocated) | sin_left_3m | Positive values for |
| | | | unaided/aided variables |
| | Speech left, | Change: | indicate speech is |
| | noise right | sin_collocated_change | louder than noise; |
| | | sin_r_change | negative indicate |
| | Noise left, | sin_l_change | speech is under the |
| | speech right | | noise |
| | | May also want change scores | |
| | | for speech to aided side and | For unilateral assigned, |
| | | speech to unaided side | also have speech to |
| | | | aided side (advantage) |
| | | | and speech to unaided side (disadvantage). |
| | | | Side (disadvalitage). |
| | | | Speech to aided |
| | | | (advantage): |
| | | | <ul> <li>If assigned R, this is</li> </ul> |
| | | | noise left, speech |
| | | | right |
| | | | right |

| | | | If assigned L, this is speech left, noise right |
|---|---|---|---|
| | | | Speech to unaided (disadvantage): If assigned R, this is speech left, noise right If assigned L, this is noise left, speech right |
| | | | Lower scores are better |
| Auditory | Unaided and | Change scores: | Continuous |
| Working<br>Memory | Aided (3 months) Recognition, | warrm_recog_change warrm_recall_change Baseline: | Sum questions 2-6 for each tasks (recognition, judgement, recall) |
| | judgement,<br>recall | warrm_recog_base warrm_recall_base warrm_judge_base | separately and get a % correct (out of 20) |
| | | 3-Months: warrm_recog_3m warrm_recall_3m warrm_judge_3m | Construct change scores as difference between 3 months and baseline for recognition and recall. |
| | | | Judgement is more of a sanity check (<90% means they probably aren't engaged) |
| | | | Higher scores are better |
| Hours of<br>Hearing Aid Use | Multiple time<br>periods (every<br>scheduled<br>visit and<br>unscheduled<br>follow ups) | Right ear: r_avg_hrs_3m r_avg_hrs_3m_na (if right HA is NA) Left ear: | How many hours on average the right/left HA was worn. NA variables: value of 1 if that HA was NA |
| | Only reporting<br>3-month<br>values here | I_avg_hrs_3m<br>I_avg_hrs_3m_na | |
| | Right and left<br>ears<br>separately | | |

# 3.2 Additional Variables of Interest

| Variable Description Variables and Source Specifications |
|----------------------------------------------------------|
|----------------------------------------------------------|

| Randomization | hearing aid | assign | Binary |
|---|---|---|---|
| assignment | assignment | | 1: unilateral 2: bilateral |
| Clinical site | Which site - | which site | Binary |
| Cirrical Site | Duke or | willen_site | 1: Vanderbilt |
| | Vanderbilt? | Character version: | 2: Duke |
| | | which_site_ch | |
| GHABP Unaided | Unaided:<br>baseline | Question 2 average, 4 standard scenarios: | For questions 2 and 3<br>(IF they answer yes to |
| | | ghabp_q2_4block_base | question 1), doing this separately by question: |
| | | Question 3 average, 4 | 4 6 1 1 1 4 |
| | | standard scenarios:<br>ghabp_q3_4block_base | 1. Subtract 1, multiply by 25, average answer to question across 4 standard scenarios |
| | | | There are 6 scenarios<br>(4 standard, 2 user-<br>nominated) |
| | | | Note that question 1 just asks if this scenario |
| | | | has happened – participants are only |
| | | | included in the |
| | | | averages if they answer "yes" |
| | | | Lower scores are better for both questions |
| ECHO | Baseline only | Global score:<br>echo_global_base | Questions 1 – 15 are used. This is scored |
| | Note: this is | | from 1-7 (or reversed |
| | the "sister" | Positive effect subscale: | for questions 2, 4, 7, |
| | questionnaire<br>to SADL | echo_positive_effect_base | 13). |
| | (aided) | Service cost subscale: | There are 4 subscales: |
| | | echo_service_cost_base | Positive Effect, Service & Cost, Negative |
| | | Negative features subscale: | Features, Personal |
| | | echo_negative_features_base | Image. For each |
| | | | subscale, the average |
| | | Personal image subscale: echo_personal_image_base | score is calculated. |
| | | | For the global score, |
| | | | this is the mean of the |
| | | | scores for all items |
| | | | (excluding question 11 if applicable). |

| TFI | Tinnitus | Voc /no. tfi. :: | Higher scores are better (higher expectations). See PCORI Scoring file for more details |
|---|---|---|---|
| | Functional Index Only at baseline | Yes/no: tfiyn Number of TFI questions missing: tfi_num_miss TFI invalid flag: tfi_invalid TFI overall score: tfi_overall_score | Non-missing if tfiyn=1 Overall score: sum all valid answers, divide by the number of questions with valid answers, multiply by 10 If more than 7 items are omitted, the overall score is not valid. 8 subscales but only reporting overall score Lower scores are better See PCORI Scoring file for more details |
| Binaural loudness summation | Baseline only CSL level right CSL level left CSL level both | binaural_r_base<br>binaural_l_base<br>binaural_both_base | Continuous |
| Dichotic digit test | Baseline only Right ear directed Left ear directed Free recall both ears Right ear free recall Left ear free recall | dichotic_r_base<br>dichotic_l_base<br>dichotic_free_both_base<br>dichotic_free_r_base<br>dichotic_free_l_base | Continuous |
| Hearing Aid<br>Fitting<br>information | Was RealEar<br>performed?<br>Which<br>WRECD was<br>used? | hafitrealear re_wrecd Ear fit Numeric: hafitwhich Character: ear_fit_ch | Yes/no for RealEar<br>performed – these<br>should all be "yes" for<br>the initial fitting |

| | Which ear was fit? | | Average/measured for WRECD – these should all be "average" at initial fitting Ear fit: 1=right 2=left 3=both |
|---|---|---|---|
| HA fit audiogram – real ear | 65 dB SPL target 65 dB SPL output UCL SPL MPO Report on differences between target and output, UCL and MPO R and L ears (may only have 1 if unilateral) 250 Hz 500 Hz 750 Hz 1000 Hz 1500 Hz 2000 Hz 3000 Hz 4000 Hz 4000 Hz 8000 Hz | Right ear: r_250_targ_out_fit r_250_ucl_mpo_fit r_500_targ_out_fit r_500_ucl_mpo_fit r_750_targ_out_fit r_750_ucl_mpo_fit r_1000_targ_out_fit r_1500_ucl_mpo_fit r_1500_ucl_mpo_fit r_1500_ucl_mpo_fit r_2000_ucl_mpo_fit r_2000_ucl_mpo_fit r_3000_ucl_mpo_fit r_3000_ucl_mpo_fit r_4000_targ_out_fit r_4000_ucl_mpo_fit r_6000_ucl_mpo_fit r_6000_ucl_mpo_fit r_8000_ucl_mpo_fit r_8000_ucl_mpo_fit l_250_ucl_mpo_fit l_500_targ_out_fit l_500_targ_out_fit l_750_targ_out_fit l_750_targ_out_fit l_750_ucl_mpo_fit l_1000_ucl_mpo_fit l_2000_ucl_mpo_fit l_2000_ucl_mpo_fit l_3000_targ_out_fit l_3000_targ_out_fit l_3000_targ_out_fit l_4000_ucl_mpo_fit l_4000_ucl_mpo_fit l_6000_targ_out_fit l_6000_ucl_mpo_fit l_6000_targ_out_fit l_6000_ucl_mpo_fit l_8000_targ_out_fit l_8000_targ_out_fit l_8000_targ_out_fit l_8000_ucl_mpo_fit | Take absolute value of the difference between target and output Take difference UCL - MPO Do plots of averages by HA configuration for each ear |

| Assigned HA 3 | 65 dB SPL | Right ear: | Take absolute value of |
|---|---|---|---|
| Month | | r_250_targ_out_3m | the difference between |
| | target | r_250_ucl_mpo_3m | |
| audiogram (real | 65 dB SPL | r_500_targ_out_3m | target and output |
| ear) | output | r_500_ucl_mpo_3m | |
| | UCL SPL | r_750_targ_out_3m | Take difference UCL - |
| | MPO | r_750_ucl_mpo_3m | MPO |
| | | r_1000_targ_out_3m | |
| | R and L ears | r_1000_ucl_mpo_3m | Do plots of averages by |
| | (may only | r_1500_targ_out_3m | HA configuration for |
| | have 1 if | r_1500_ucl_mpo_3m | each ear |
| | unilateral) | r_2000_targ_out_3m | |
| | | r_2000_ucl_mpo_3m | |
| | 250 Hz | r_3000_targ_out_3m | |
| | 500 Hz | r_3000_ucl_mpo_3m | |
| | 750 Hz | r_4000_targ_out_3m | |
| | 1000 Hz | r_4000_ucl_mpo_3m | |
| | 1500 Hz | r_6000_targ_out_3m | |
| | 2000 Hz | r_6000_ucl_mpo_3m | |
| | | r_8000_targ_out_3m | |
| | 3000 Hz | r_8000_ucl_mpo_3m | |
| | 4000 Hz | | |
| | 6000 Hz | | |
| | 8000 Hz | Left ear: | |
| | | I_250_targ_out_3m | |
| | | l_250_ucl_mpo_3m | |
| | | I_500_targ_out_3m | |
| | | I_500_ucl_mpo_3m | |
| | | I_750_targ_out_3m | |
| | | I_750_ucl_mpo_3m | |
| | | I_1000_targ_out_3m | |
| | | l_1000_ucl_mpo_3m | |
| | | I_1500_targ_out_3m | |
| | | l_1500_ucl_mpo_3m | |
| | | I_2000_targ_out_3m | |
| | | l_2000_ucl_mpo_3m | |
| | | I_3000_targ_out_3m | |
| | | l_3000_ucl_mpo_3m | |
| | | I_4000_targ_out_3m | |
| | | l_4000_ucl_mpo_3m | |
| | | I_6000_targ_out_3m | |
| | | l_6000_ucl_mpo_3m | |
| | | I_8000_targ_out_3m | |
| | | l_8000_ucl_mpo_3m | |

# 4 Statistical Analysis Plan

Analysis: To be completed by December 31, 2024.

### 4.1 Aim: compare all outcomes between the two arms

Compare the outcomes between the two arms (bilateral hearing aid and unilateral hearing aid) at 3 months.

**Analysis:** This will be reported for patients who have 3-month scores ("completers"). The primary analysis will be performed using either t-tests or Kruskal Wallis tests depending on whether or not the outcome

distributions appear to be normally distributed. The total score for each survey at 3 months or the benefit score will be used as the outcomes. For GHABP, we will compare the four standard questions (averaged and standardized) for the 4 standard scenarios between the two arms at 3 months for patients who answer "yes" to the first question (if the scenario happens).

The null hypothesis is that the means of the outcomes for the two treatment groups are the same.

 $H_0$ :  $\mu_{unilateral} = \mu_{bilateral}$ 

| | Unilateral (N=XXX) | Bilateral (N=XXX) | P-Value* |
|---|---|---|---|
| GHABP Aided: In this situation, | | | |
| what proportion of the time do | | | XXX |
| you wear your hearing aid? | | | |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| GHABP Aided: In this situation, | | | |
| how much does your hearing aid | | | XXX |
| help you? | | | |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| GHABP Aided: In this situation, | | | |
| with your hearing aid, how much | | | XXX |
| difficulty do you now have? | | | |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| GHABP Aided: For this situation, | | | |
| how satisfied are you with your | | | XXX |
| hearing aid? | | | |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| SADL Global Score | | | XXX |
| N | XXX | XXX | |

| Missing | XXX | XXX | |
|-----------------------------------------|-----------|-----------|-----|
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| HHI-E Change Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| IOI-HA Total Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| SSQ Change Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| Speech and Noise Test: 0 Degrees | | | WW |
| (Co-located) Change Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| Auditory Working Memory - | | | WW |
| Recognition Change Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| <b>Auditory Working Memory - Recall</b> | | | |
| Change Score | | | |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |

We will create boxplots or other figures displaying the distributions of these outcomes by randomization. These figures may supplement or replace Table 1 above.

### 4.2 Aim: descriptive tables/plots for additional variables

Analysis: we will describe or plot the distributions of additional variables at baseline, hearing aid fit, or 3 month visit as appropriate by assigned treatment. For GHABP, the two unaided (baseline) questions and the one aided (3-month) question (averaged and standardized) will only include patients who answered "yes" to the first question (if the scenario happens). These will be reported across the 4 standard scenarios.

| | Unilateral (N=XXX) | Bilateral (N=XXX) |
|--------------------------------|--------------------|-------------------|
| GHABP Unaided: How much | | |
| difficulty do you have in this | | |
| ituation? | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| GHABP Unaided: How much | | |
| loes any difficulty in this | | |
| ituation worry, annoy or up | set | |
| ou? | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| with your hearing aid, how | | |
|---|---|---|
| much does any difficulty in this | | |
| - | | |
| situation worry, annoy, or upset | | |
| you? | XXX | XXX |
| N<br>Missing | XXX | XXX |
| Missing | | |
| Mean (SD)<br>Median | XXX (XXX)<br>XXX | XXX (XXX)<br>XXX |
| Q1, Q3 | XXX, XXX<br>XXX - XXX | XXX, XXX<br>XXX - XXX |
| Range | ^^^ - ^^^ | \\\\ - \\\\ |
| ECHO Global Score (Baseline) | XXX | XXX |
| N<br>Missing | | |
| Missing | XXX | XXX |
| Mean (SD)<br>Median | XXX (XXX) | XXX (XXX) |
| | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| ECHO Positive Effect Subscale | | |
| (Baseline) | VVV | VVV |
| N<br>Missing | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| ECHO Service Cost Subscale | | |
| (Baseline) | VVV | VVV |
| N<br>Missing | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| ECHO Negative Features | | |
| Subscale (Baseline) N | VVV | VVV |
| | XXX<br>XXX | XXX<br>XXX |
| Missing | XXX (XXX) | |
| Mean (SD)<br>Median | XXX | XXX (XXX) |
| | | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX<br>XXX - XXX |
| Range | XXX - XXX | \\\\ - \\\\ |
| ECHO Personal Image Subscale | | |
| (Baseline) | VVV | VVV |
| N<br>Missing | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD)<br>Median | XXX (XXX) | XXX (XXX) |
| | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |

**GHABP Aided: In this situation,** 

| SADL Positive Effect Subscale (3 | | |
|----------------------------------|-----------|-----------|
| Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SADL Service Cost Subscale (3 | | |
| Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SADL Negative Features | | |
| Subscale (3 Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SADL Personal Image Subscale (3 | | |
| Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| HHI-E Total Score (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| HHI-E Total Score (3-Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| HHI-E Situational Subscale | | |
| (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |

| | | , . |
|--------------------------------|------------|------------|
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| HHI-E Situational Subscale (3- | | |
| Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| HHI-E Emotional Subscale | | |
| (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| HHI-E Emotional Subscale (3- | | |
| Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Tinnitus Presence (Baseline) | | |
| No | XXX (XXX%) | XXX (XXX%) |
| Yes | XXX (XXX%) | XXX (XXX%) |
| Missing | XXX (XXX%) | XXX (XXX%) |
| TFI Overall Score (Baseline) | | |
| N | XXX | XXX |
| Not Applicable (Answered No | XXX | XXX |
| to Presence) | | |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Overall Score (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Overall Score (3-Month) | | |
| N | XXX | XXX |

| Missing | XXX | XXX |
|----------------------------------|--------------|-----------|
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX, XXX | XXX, XXX |
| SSQ Speech/Hearing Subscale | | 7000 7000 |
| (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Speech/Hearing Subscale | | |
| (3-Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | xxx | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Spatial/Hearing Subscale | | |
| (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Spatial/Hearing Subscale (3- | | |
| Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Qualities of Hearing | | |
| Subscale (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Qualities of Hearing | | |
| Subscale (3-Month) | <b>100</b> / | 1007 |
| N<br>Mississe | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |

| No. dia | VVV | V/// |
|---|---|---|
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Binaural Loudness Summation: | | |
| Right (Baseline) N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX, XXX |
| Binaural Loudness Summation: | XXX XXX | 7000 7000 |
| Left (Baseline) | | |
| N N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Binaural Loudness Summation: | | |
| Both (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Dichotic Digits: Right Ear | | |
| Directed (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Dichotic Digits: Left Ear Directed | | |
| (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Dichotic Digits: Free Recall Both | | |
| (Baseline)<br>N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Q1, Q0 | 700,700 | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |

| Range | XXX - XXX | XXX - XXX |
|---|---|---|
| Dichotic Digits: Free Recall Right | ^^^ - ^^^ | \\\\ - \\\\ |
| (Baseline) | | |
| N | XXX | XXX |
| | XXX | XXX |
| Missing | | |
| Mean (SD)<br>Median | XXX (XXX)<br>XXX | XXX (XXX)<br>XXX |
| Q1, Q3 | XXX, XXX<br>XXX - XXX | XXX, XXX<br>XXX - XXX |
| Range | *** - *** | XXX - XXX |
| Dichotic Digits: Free Recall Left | | |
| (Baseline) | VVV | VVV |
| N<br>Missing | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX<br>XXX - XXX |
| Range | XXX - XXX | XXX - XXX |
| Speech and Noise Test: 0 | | |
| Degrees (Co-located) Score (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Speech and Noise Test: 0 | XXX - XXX | \\\\ - \\\\\ |
| Degrees (Co-located) Score (3- | | |
| Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Speech and Noise Test: Speech | 700. | 7000 7000 |
| Left, Noise Right Score | | |
| (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | xxx | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Speech and Noise Test: Speech | | |
| Left, Noise Right Score (3- | | |
| Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| | • • | , , |

| Median | XXX | XXX |
|---------------------------------|-----------|-------------|
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Speech and Noise Test: Speech | XXX - XXX | XXX - XXX |
| Left, Noise Right Change Score | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Speech and Noise Test: Noise | | 7000 7000 |
| Left, Speech Right Score | | |
| (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | xxx | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Speech and Noise Test: Noise | | |
| Left, Speech Right Score (3- | | |
| Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Speech and Noise Test: Noise | | |
| Left, Speech Right Change Score | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Auditory Working Memory - | | |
| Recognition Score (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Auditory Working Memory - | | |
| Recognition Score (3-Month) | NAA/ | <b>1777</b> |
| N<br>Missing | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |

| Median | xxx | XXX |
|----------------------------|-----------|-----------|
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Auditory Working Memory - | | |
| Recall Score (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Auditory Working Memory - | | |
| Recall Score (3-Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Auditory Working Memory - | | |
| Judgement Score (Baseline) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Auditory Working Memory - | | |
| Judgement Score (3-Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |

We will plot the average absolute difference between target and output at each frequency for each ear by assigned hearing aid configuration for both the hearing aid fit and 3-month visits (with visits either grouped together in the same plot or plotted separately). We will also do this for the average difference between MPO and UCL at each frequency.

#### 5 Future Plans

There are additional items we may wish to explore in the future, at which point a new SAP will be developed. Ideas include looking at:

- Additional GHABP measures
- EMA surveys
- Mask questions

- Additional hearing aid hours of use Unscheduled visits

## Statistical Analysis Plan (SAP) – Secondary (6-Month) Outcomes and Descriptives

Project: Evaluation of Unilateral vs Bilateral Hearing Aids for the Treatment of Age-related Hearing

Loss

IRB Number: Pro00106077

Investigator(s): Sherri Smith, AuD, PhD

Biostatisticians: Rebecca North, PhD, Kayla Kilpatrick, PhD, Sarah Peskoe, PhD, Frank Rockhold, PhD

**Original Creation Date:** 01.07.2025

Version Date: 01.07.2025

| Investigator Agreement | <ul> <li>□ All statistical analyses included in an abstract or manuscript should reflect the work of the biostatistician(s) listed on this SAP. No changes or additional analyses should be made to the results or findings without discussing with the project biostatistician(s).</li> <li>□ All biostatisticians on this SAP should be given sufficient time to review the full presentation, abstract, manuscript, or grant and be included as co-authors on any abstract or manuscript resulting from the analyses.</li> <li>□ If substantial additional analysis is necessary or the aims of the project change, a new SAP will need to be developed.</li> <li>□ Publications resulting from this SAP are supported in part by the Duke CTSA and must cite grant number UL1TR002553 and be submitted to PubMed Central.</li> <li>□ I have reviewed the SAP and understand that any changes must be documented.</li> </ul> Acknowledged by: Click or tap here to enter text. |
|---|---|
| | Date: Click or tap to enter a date. |
| | Dute. of tap to effect a dute. |

#### **Activity Log**

| Acronyms | APHAB | Abbreviated Profile of Hearing Aid Benefit |
|----------|--------|---------------------------------------------------|
| | IOI-HA | International Outcomes Inventory for Hearing Aids |
| | SADL | Satisfaction with Amplification in Daily Life |
| | SSQ | Speech Spatial Qualities |
| | HHIE | Hearing Handicap Inventory for Elderly |

# 1 Study Overview

Background/Introduction: The overall goal of the project is to determine the benefit of unilateral or bilateral hearing aid fittings in adults with mild-to-moderate age-related hearing loss. This will address the lack of high-quality evidence supporting bilateral hearing aids over unilateral hearing aids. This project will use a randomized controlled trial with two treatment arms: a bilateral hearing aid fitting group and a unilateral hearing aid fitting group.

#### 1.1 Aims for Secondary Outcomes

- Compare all outcomes between the two arms (bilateral hearing aid and unilateral hearing aid) at 6 months. The primary hypothesis is that bilateral hearing aids are superior to the unilateral hearing aids with respect to the overall patient-reported benefit.
  - o Descriptive tables for additional clinical variables at 6-months by assigned treatment
  - Plots of APHAB Global score and change from baseline by assigned treatment
- Compare all outcomes at 6 months by final configuration choice
- Compare all outcomes at 6 months by switching status relative to baseline

# 2 Study Population

#### 2.1 Inclusion Criteria

- 50+ years of age
- Mild to moderate, symmetrical SNHL (symmetrical: < 20 dB between ears on average from 500-4000 Hz)
- Open-mindedness to unilateral or bilateral amplification
- No prior hearing aid experience
- Adequate literacy to complete questionnaires
- Willing to purchase study-specific hearing aid(s)

#### 2.2 Exclusion Criteria

- Concerns for middle ear pathology
- Concerns for retrocochlear pathology
- Severe tinnitus as the reason for seeking amplification
- Co-morbid condition that would interfere with study (e.g., dementia, blindness, neurologic pathology)
- History of fluctuating hearing loss

#### 2.3 Data Acquisition

Fill in all relevant information:

| Study design | Randomized controlled trial with 2 arms (bilateral hearing aid, unilateral hearing aid) |
|---|---|
| | Note: Randomization was stratified by clinical site. |
| Data source/how the data were collected | Screening information pulled from EHR data |
| | Baseline surveys captured via in-person interview and |
| | recorded in REDCap |
| Contact information for team member | All data access is through |
| responsible for data | . Questions on data validity |
| collection/acquisition | will go to PI: Sherri Smith (Sherri.smith@duke.edu) |
| Date or version (if downloaded, provide | 10.28.2024 |
| date) | |
| Data transfer method and date | Direct data extraction from REDCap |
| Where dataset is stored | REDCap |
| | Extracted data and analytic datasets are stored on a |
| | secure drive in the CRU folder: \\duhs-vclin- |
| | <pre>nc1\dusom biostats fs\Data\BiostatsCore\CRU\Head</pre> |
| | and Neck\Smith\PCORI Pro00106077\Data pulls |

Notes: Additional variable details for all variables can be found in the "PCORI Variable Details" Excel file. Scoring details can be found in "PCORI Scoring 20240923".

# 3 Outcomes, Exposures, and Additional Variables of Interest

### 3.1 Outcome(s)

| Outcome | Description | Variables and Source | Specifications |
|---|---|---|---|
| APHAB<br>Change<br>Score | Difference in aided APHAB scores at month 6 and unaided scores at baseline | aphab_global_change_6m (constructed in analytic script) | Scale score – will need to calculate global communication scores at baseline (unaided) and 3 months (aided), subtract (3 months – baseline) A lower score on APHAB is better. Rescore variables and multiply by 100 1 = 0.99 2 = 0.87 3 = 0.75 4 = 0.50 5 = 0.25 6 = 0.12 7 = 0.01 Reverse score questions 1, 9, 11, 16, 19, 21 Global score: mean of variables in the EC, BN, RV subscale scores (excludes questions 3, 8, 13, 17, 20, 22) Note: APHAB has 4 subscales and a global communication scale. The study is powered based on the benefit score on the global communication scale (August 2019 draft – APHAB SD of 25 with different |
| APHAB<br>change | Responders vs non- | Decrease of 25 units:<br>aphab responder25 6m | levels of Cohen's D). Patients with a decrease of at least 25 units (or 15 units for |
| score –<br>binary, 6<br>months | responders<br>for primary<br>APHAB<br>outcome | Decrease of 15 units: aphab_responder15_6m (Constructed in analytic script) | the sensitivity analysis) on the APHAB scale at month 6 will be considered "responders." Patients not returning or who do not have a score at 6 |

| | | | months will be considered "non-responders." Patients with a baseline score < 25 (or < 15) are ineligible (missing). Binary (25 unit decrease): Missing if baseline score <25 1 if aphab_global_change_6m <=-25 0 else Binary (15 unit decrease); Missing if baseline score <15 1 if aphab_global_change_6m <=-15 0 else |
|---|---|---|---|
| APHAB – 4 subscales | EC, BN, RV, AV scales at 6 months and change score relative to baseline | 6-month variables: aphab_ec_6m aphab_bn_6m aphab_rv_6m aphab_av_6m | Rescore variables and multiply by 100 1 = 0.99 2 = 0.87 3 = 0.75 4 = 0.50 5 = 0.25 6 = 0.12 7 = 0.01 Reverse score questions 1, 9, 11, 16, 19, 21 EC: mean of questions 4, 10, 12, 14, 15, 23 BN: mean of questions 1, 6, 7, 16, 19, 24 RV: mean of questions 2, 5, 9, 11, 18, 21 AV: mean of questions 3, 8, 13, 17, 20, 22 |
| IOI-HA | Total score<br>Note: this is<br>measured<br>only at 3 and<br>6 months | ioiha_total_6m | Total score: sum responses to questions 1-7 (should be on a range between 1-5). Item 8 is self-perceived hearing difficulty used for normative purposes (currently not used as part of total score) |

| | | | This is initially coded as 0 to 4 in REDCap – changed to 1-5 Currently, we're treating IOI-HA total score as continuous, but this may need to be treated as ordinal. |
|---|---|---|---|
| SADL | Note: this is measured | Global score: sadl_global_6m | Higher scores are better Questions 1 – 15 are used. This is scored from 1-7 (or reversed |
| | only at 3 and 6 months. | Positive effect subscale: sadl_positive_effect_6m | for questions 2, 4, 7, 13). |
| | Note: the "sister" questionnaire at baseline is ECHO | Service cost subscale: sadl_service_cost_6m Negative features subscale: sadl_negative_features_6m | There are 4 subscales: Positive Effect, Service & Cost, Negative Features, Personal Image. For each subscale, the average score is calculated. |
| | | Personal image subscale: sadl_personal_image_6m | For the global score, this is the mean of the scores for all items (excluding questions 11 and 14 if applicable). |
| | | | Higher scores are better (higher satisfaction). |
| | | | See PCORI Scoring file for more details |
| SSQ | Note: this is<br>measured at<br>baseline, 3<br>months, and<br>6 months. | Change score (constructed in analytic script): ssq_overall_change_6m Baseline: Overall score: ssq_overall_base | 3 subscales: Speech is questions 1 – 14 (corresponds to the "pt1" variables). Spatial is 17 questions (corresponds to the "pt2" variables). Qualities is 18 questions (correspond to the "pt3" variables). |
| | | Speech/hearing subscale: ssq_speech_hearing_base | Overall score: mean of the items. |
| | | Spatial/hearing subscale: ssq_spatial_hearing_base | For instances where people mark NA and a value, if the value is 50, set as NA. If a value |
| | | Qualities of hearing subscale: ssq_qualities_of_hearing_base | other than 50, use that value. |
| | | 6-Months: Overall score: ssq_overall_6m | We will also create a change score as the difference in the overall score between 6 months and baseline (6 months – baseline) |

| | | Speech/hearing subscale: | |
|---|---|---|---|
| | | ssq_speech_hearing_6m | Higher scores are better |
| | | Spatial/hearing subscale: | |
| | | ssq_spatial_hearing_6m | |
| | | Qualities of hearing subscale: | |
| | | ssq_qualities_of_hearing_6m | |
| HHI-E | Note: this is | Change score (constructed in | Yes = 4 points, Sometimes = 2 |
| | measured at | analytic script): | points, and No = 0 points. |
| | baseline, 3 months, and | hhie_total_change_6m | Total scale score = sum of all |
| | 6 months | Baseline: | 25 items |
| | | Total score: hhie_total_base | |
| | | C : 1/C': .: | Social/Situational subscale: |
| | | Social/Situational subscale: hhie_situational_base | questions 1, 3, 6, 8, 10, 11 13, 15, 16, 19, 21, 23 |
| | | Emotional subscale: | Emotional subscale: questions |
| | | hhie_emotional_base | 2, 4, 5, 7, 9, 12, 14, 17, 18, 20, 22, 24, 25 |
| | | 6-Months: | , , |
| | | Total score: hhie_total_6m | We will also create a change score as the difference in the |
| | | Social/Situational subscale: | total scale score between 6 |
| | | hhie_situational_6m | months and baseline (6 |
| | | Emotional subscale: | months – baseline) |
| | | hhie_emotional_6m | Lower scores are better |

# 3.2 Additional Variables of Interest

| Variable | Description | Variables and Source | Specifications |
|---|---|---|---|
| Randomization | hearing aid | assign | Binary |
| assignment | assignment | | 1: unilateral |
| | | | 2: bilateral |
| Clinical site | Which site - | which_site | Binary |
| | Duke or | | 1: Vanderbilt |
| | Vanderbilt? | Character version: | 2: Duke |
| | | which_site_ch | |
| Switch | Patients are | ha_switch_assign_6m | Binary: |
| configuration at 6 | given the | | 1: Switched |
| months | opportunity | | configuration |
| | to switch | | 0: Didn't switch |
| | configuration | | |
| | at 3 months | | Switched configuration |
| | and make a | | is defined as unilateral |
| | final | | to bilateral or vice |
| | configuration | | versa (do not count |

| | choice at 6<br>months | | switching unilateral to<br>a different ear as a<br>switch) |
|---|---|---|---|
| | | | Switched configuration also includes switching from 1 or 2 to 0 |
| 6-month final choice configuration | Patients are given to opportunity to make a final choice of hearing aid configuration at 6 months | ha_final_choice_6m Character version: ha_final_choice_6m_ch | Categorical: Right Left Both None Missing |

# 4 Statistical Analysis Plan

Deadline: To be completed by January 24, 2025.

#### 4.1 Aim: compare all outcomes between the two assigned treatment arms

Compare the outcomes between the two assigned treatment arms (bilateral hearing aid and unilateral hearing aid) at 6 months.

Analysis: This will be reported for patients who have 6-month scores ("completers"). The analysis will be performed using either t-tests or Kruskal Wallis tests depending on whether or not the outcome distributions appear to be normally distributed for continuous outcomes. The total score for each survey at 6 months or the benefit score will be used as the outcomes. The Chi-Square test will be used for the APHAB Responder outcomes, with patient counts and relative frequencies reported.

The null hypothesis is that the means of the outcomes for the two treatment groups are the same.

 $H_0$ :  $\mu_{unilateral} = \mu_{bilateral}$ 

| | Unilateral (N=XXX) | Bilateral (N=XXX) | P-Value* |
|---|---|---|---|
| APHAB Global Change Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| APHAB Responder (25 Units)** | | | XXX |
| No | XXX (%) | XXX (%) | |
| Yes | XXX (%) | XXX (%) | |
| Ineligible to Drop 25 Units | XXX | XXX | |
| APHAB Responder (15 Units)** | | | XXX |
| No | XXX (%) | XXX (%) | |
| Yes | XXX (%) | XXX (%) | |
| | 10 W | | Page |

| Ineligible to Drop 15 Units | XXX | XXX | |
|-----------------------------|-----------|-----------|-----|
| SADL Global Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| HHI-E Change Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| IOI-HA Total Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |
| SSQ Change Score | | | XXX |
| N | XXX | XXX | |
| Missing | XXX | XXX | |
| Mean (SD) | XXX (XXX) | XXX (XXX) | |
| Median | XXX | XXX | |
| Q1, Q3 | XXX, XXX | XXX, XXX | |
| Range | XXX - XXX | XXX - XXX | |

<sup>\*</sup>T-test/Kruskal Wallis or Chi-Square test

We will also describe the distributions of additional variables at 6-month visit as appropriate by assigned treatment (subscales and total scores where change score was reported above). We will also create boxplots for APHAB Global total score and change score by randomization. These figures may supplement Table 1 above.

| | Unilateral (N=XXX) | Bilateral (N=XXX) |
|----------------------------|--------------------|-------------------|
| APHAB Global Total Score ( | 5 | |
| Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| APHAB EC Subscale (6 Mont | :hs) | |
| N | XXX | XXX |
| Missing | XXX | XXX |

<sup>\*\*</sup>Denominator for percentages does not include patients ineligible to drop 'x' units

| Maan (CD) | VVV (VVV) | VVV (VVV) |
|--------------------------------|------------------|------------------|
| Mean (SD)<br>Median | XXX (XXX)<br>XXX | XXX (XXX)<br>XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| APHAB EC Subscale Change Score | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| APHAB BN Subscale (6 Months) | 7001 | 7000 7000 |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | xxx | XXX |
| Q1, Q3 | xxx, xxx | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| APHAB BN Subscale Change Score | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| APHAB RV Subscale (6 Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| APHAB RV Subscale Change Score | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| APHAB AV Subscale (6 Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| APHAB AV Subscale Change Score | MAX | <b>3337</b> |
| N<br>Missing | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |

| Median | XXX | XXX |
|-----------------------------------|-----------|-------------|
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SADL Positive Effect Subscale (6 | AAA - AAA | //// - //// |
| Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SADL Service Cost Subscale (6 | | 7000 7000 |
| Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | xxx | XXX |
| Q1, Q3 | xxx, xxx | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SADL Negative Features Subscale | | |
| (6 Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SADL Personal Image Subscale (6 | | |
| Months) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| HHI-E Total Score (6-Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| HHI-E Social/Situational Subscale | | |
| (6-Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |

| HHI-E Emotional Subscale (6- | | |
|-----------------------------------|-----------|-----------|
| Month) | VVV | WW |
| N<br>Minain a | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Overall Score (6-Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Speech/Hearing Subscale (6- | | |
| Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Spatial/Hearing Subscale (6- | | |
| Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| SSQ Qualities of Hearing Subscale | | |
| (6-Month) | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | xxx | xxx |
| Q1, Q3 | XXX, XXX | xxx, xxx |
| Range | XXX - XXX | XXX - XXX |

### 4.2 Aim: Compare 6-month outcomes by 6-month final choice of HA configuration

Compare the outcomes between the two HA configuration choice groups (bilateral hearing aid and unilateral hearing aid) at 6 months.

**Analysis:** Similar analysis and table as in Aim 1, Table 1, but with columns defined by 6-month HA configuration choice [Table 3].

#### 4.3 Aim: Compare 6-month outcomes by 6-month configuration switching status relative to baseline

Compare the outcomes between the two groups (switched or did not switch from assigned HA configuration) at 6 months.

**Analysis:** Similar analysis and table as in Aim 1, Table 1, but with columns defined by 6-month HA switching status relative to baseline [Table 4].

#### 4.4 Initially planned analyses that we will not do

We had initially planned to estimate repeated measures mixed models for all outcomes gathered at baseline, 3-months, and 6-months with randomized treatment assignment as the covariate of interest. However, given the propensity for participants to switch hearing aid configurations at 3-months and that there are only 2 follow-up timepoints, we deemed it more appropriate to look at the outcomes cross-sectionally rather than longitudinally.

#### 5 Future Plans

There are additional items we may wish to explore in the future, at which point a new SAP will be developed. Ideas include looking at:

- Additional Glasgow Hearing Aid Benefit Profile measures
- Mask questions
- · Additional hearing aid hours of use
- Unscheduled visits

## Statistical Analysis Plan (SAP) – EMAs

**Project:** Evaluation of Unilateral vs Bilateral Hearing Aids for the Treatment of Age-related Hearing Loss **IRB Number:** Pro00106077 Investigator(s): Sherri Smith, AuD, PhD Biostatisticians: **Original Creation Date: 02.18.2022** Version Date: 12.02.2024 ☐ All statistical analyses included in an abstract or manuscript should **Investigator Agreement** reflect the work of the biostatistician(s) listed on this SAP. No changes or additional analyses should be made to the results or findings without discussing with the project biostatistician(s). ☐ All biostatisticians on this SAP should be given sufficient time to review the full presentation, abstract, manuscript, or grant and be included as co-authors on any abstract or manuscript resulting from the analyses. ☐ If substantial additional analysis is necessary or the aims of the project change, a new SAP will need to be developed. ☐ Publications resulting from this SAP are supported in part by the Duke CTSA and must cite grant number UL1TR002553 and be submitted to PubMed Central. □ I have reviewed the SAP and understand that any changes must be documented. Acknowledged by: Click or tap here to enter text. Date: Click or tap to enter a date. 02.18.2022 Created SAP for GHABP and EMA outcomes **Activity Log** 02.21.2022 Added details to analysis 03.14.2022 Updated based on discussion 01.26.2023 Add additional details to variables and updates reflective of changes made in other SAPs 05.31.2024 Moved 6-month data to Future Plans section 12.02.2024 Removed GHABP and moved user-nominated scenarios to Future Plans section APHAB Abbreviated Profile of Hearing Aid Benefit Acronyms **EMA Ecological Momentary Assessment GHABP** Glasgow Hearing Aid Benefit Profile IOI-HA International Outcomes Inventory for Hearing Aids SADL Satisfaction with Amplification in Daily Life SSQ Speech Spatial Qualities Hearing Handicap Inventory for Elderly HHIE

## 1 Study Overview

Background/Introduction: The overall goal of the project is to determine the benefit of unilateral or bilateral hearing aid fittings in adults with mild-to-moderate age-related hearing loss. This will address the lack of high-quality evidence supporting bilateral hearing aids over unilateral hearing aids. This project will use a randomized controlled trial with two treatment arms: a bilateral hearing aid fitting group and a unilateral hearing aid fitting group.

#### 1.1 Aim

 Compare EMA outcome between the two arms across all responses to the 4 standard scenarios, looking at the time periods from baseline to 3 months and 3 months to 6 months.

# 2 Study Population

#### 2.1 Inclusion Criteria

- 50+ years of age
- Mild to moderate, symmetrical SNHL (symmetrical: < 20 dB between ears on average from 500-4000 Hz)
- Open-mindedness to unilateral or bilateral amplification
- No prior hearing aid experience
- Adequate literacy to complete questionnaires
- Willing to purchase study-specific hearing aid(s)

#### 2.2 Exclusion Criteria

- Concerns for middle ear pathology
- Concerns for retrocochlear pathology
- Severe tinnitus as the reason for seeking amplification
- Co-morbid condition that would interfere with study (e.g., dementia, blindness, neurologic pathology)
- History of fluctuating hearing loss

#### 2.3 Data Acquisition

#### Fill in all relevant information:

| Study design | Randomized controlled trial with 2 arms (bilateral hearing aid, unilateral hearing aid) |
|---|---|
| | Note: Randomization was stratified by clinical site. |
| Data source/how the data were collected | Screening information pulled from EHR data |
| | Baseline surveys captured via in-person interview and recorded in REDCap |
| Contact information for team member | All data access is through |
| responsible for data | . Questions on data validity |
| collection/acquisition | will go to PI: Sherri Smith (Sherri.smith@duke.edu) |
| Date or version (if downloaded, provide | 10.17.2024 |
| date) | |
| Data transfer method and date | Direct data extraction from REDCap |
| Where dataset is stored | REDCap |
| | Extracted data and analytic datasets are stored on a |
| | secure drive in the CRU folder: \\duhs-vclin- |

# 3 Outcomes, Exposures, and Additional Variables of Interest

# 3.1 Outcome(s)

| Outcome | Description | Variables and Source | Specifications |
|---|---|---|---|
| GHABP Unaided | GHABP is<br>measured at<br>baseline<br>(unaided) | GHABP unaided: ghabun1a – ghabun6c 3 total questions for each of 6 scenarios (4 standard, 2 user- nominated) First question just asks if this scenario has happened – ONLY include those who say yes to this | For questions 2 and 3 (IF they answer yes to question 1), doing this separately by question: 1. Subtract 1, multiply by 25, average answer to question across 4 standard scenarios 2. Subtract 1, multiply by 25, average answer to question across 2 user-nominated scenarios 3. Subtract 1, multiply by 25, average answer to question across all 6 scenarios. For self-nominated goals, people may write in "NA", "N/A", "Na", "None", "Not applicable" – these should |
| GHABP Aided | GHABP is<br>measured at 3<br>months<br>(aided) | GHABP aided: ghaba1a_v1 – ghaba6f_v1 6 total questions for each of 6 scenarios (4 standard, 2 user- nominated) First question just asks if this scenario has happened – ONLY include those who say yes to this | be ignored (set to missing) For questions 3-6 (IF they answer yes to question 1), doing this separately by question: 1. Subtract 1, multiply by 25, average answer to question across 4 standard scenarios 2. Subtract 1, multiply by 25, average answer to question across 2 user-nominated scenarios 3. Subtract 1, multiply by 25, average answer to question across all 6 scenarios. Note: ignore current question 2 as it is non-standard |

| | | | For self-nominated goals, people may write in "NA", "N/A", "Na", "None", "Not applicable" – these should be ignored (set to missing). Note: we will need to keep track of these baseline goals in case people answer "yes" at the later timepoints. |
|---|---|---|---|
| EMA | EMA are surveys (same questions as GHABP) sent 5 times a day for a week. Have these in two time periods: before 3 months and after 3 months. These time periods will be kept separate. | EMA variables: for Duke, these are ghaba1a – ghaba6f. For Vanderbilt, these are ghaba1a_v2 – ghaba6f_v2. Have EMA "events" EMA 1a – EMA 7e for survey before 3 months. Have EMA "events" EMA 8a – EMA 14e for surveys after 3 months (before 6 months) 6 total questions for each of 6 scenarios (4 standard, 2 user- nominated) First question just asks if this scenario has happened – ONLY include those who say yes to this | Several pieces here. First, for questions 3-6 (IF they answer yes to question 1), subtract 1 and multiply by 25. Then interested in 2 cases: 1. Look at answer to all question X's over ALL scenarios for blocks of scenarios below 2. For question X, look at answer to all question X's within a given scenario for the 4 standard scenarios Blocks of scenarios: 1. 4 standard scenarios 2. 2 user-nominated scenarios 3. All 6 scenarios. Note: ignore current question 2 as it is non-standard For self-nominated goals, people may write in "NA", "N/A", "Na", "None", "Not applicable" – these should be ignored (set to missing). Note: we will need to keep track of these baseline goals in case people answer "yes" at the later timepoints. |

Notes: 6 total scenarios, 4 standard, 2 user-nominated. Standard scenarios:

- 1. LISTENING TO THE TELEVISION WITH OTHER FAMILY OR FRIENDS WHEN THE VOLUME IS ADJUSTED TO SUIT OTHER PEOPLE
- 2. HAVING A CONVERSATION WITH ONE OTHER PERSON WHEN THERE IS NO BACKGROUND NOISE

- 3. CARRYING ON A CONVERSATION IN A BUSY STREET OR SHOP
- 4. HAVING A CONVERSATION WITH SEVERAL PEOPLE IN A GROUP

#### Unaided questions:

- 1. Does this situation happen in your life?
- 2. How much difficulty do you have in this situation?
- 3. How much does any difficulty in this situation worry, annoy or upset you?

#### Aided/EMA questions:

- 1. Did this situation happen in the past few weeks? (GHABP aided) OR Did this situation happen in the last three hours? (EMA)
- 2. In this situation, with your hearing aid, how much does any difficulty in this situation worry, annoy or upset you? (NOTE: ignore this question as it is non-standard)
- 3. In this situation, what proportion of the time do you wear your hearing aid?
- 4. In this situation, how much does your hearing aid help you?
- 5. In this situation, with your hearing aid, how much difficulty do you now have?
- 6. For this situation, how satisfied are you with your hearing aid?

#### 3.2 Additional Variables of Interest

| Variable | Description | Variables and Source | Specifications |
|---------------|--------------|------------------------|----------------|
| Randomization | hearing aid | Baseline visit: assign | Binary |
| assignment | assignment | | 1: unilateral |
| | | | 2: bilateral |
| Clinical site | Which site - | Baseline visit: | Binary |
| | Duke or | which_site | 1: Vanderbilt |
| | Vanderbilt? | | 2: Duke |

# 4 Statistical Analysis Plan

Analysis: To be completed by December 31, 2024

#### 4.1 Descriptive Characteristics for EMA Surveys

Analysis: We will present the mean with standard deviation (SD), median with interquartile range (IQR), and ranges (min and max) for number of EMA surveys completed. The 0-3-month period and 3-6-month period will be done separately, stratified by baseline assignment and 3M choice, respectively.

| Table 1: EMA Summaries | | |
|---|---|---|
| Number of EMA Surveys Completed<br>Before 3 Months | Assigned Unilateral (N=XXX) | Assigned Bilateral (N=XXX) |
| N | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |
| Number of EMA Surveys Completed | 3M Choice – Unilateral | 3M Choice – Bilateral |
| After 3 Months | (N=XXX) | (N=XXX) |
| N | XXX | XXX |

| Mean (SD) | XXX (XXX) | XXX (XXX) |
|-----------|-----------|-----------|
| Median | XXX | XXX |
| Q1, Q3 | XXX, XXX | XXX, XXX |
| Range | XXX - XXX | XXX - XXX |

# 4.2 Aim: compare EMA surveys between the two arms in the period between baseline and 3 months, and between 3M choice groups between 3 months and 6 months

For question X, we want to look at the answers to all question X's over the 4 standard scenarios.

Analysis: This will be done using intent-to-treat for patients who have EMA surveys and answer "yes" to the first question (if the scenario happens). The primary analysis will be performed by linear mixed effects models with covariates clinical site and assigned treatment/3M choice, with a separate model for each question. The overall average of within-person means will be reported by treatment arm/3M choice, as well as T-test p-values from the fitted models for the treatment arm/3M choice covariate, where a p-value < 0.05 would indicate a difference in average response between treatment arms/3M choices.

| Question & Scenarios | Assigned Unilateral | Assigned Bilateral | P-Value <sup>3</sup> |
|---|---|---|---|
| 0-3 Months | (Overall Mean) | (Overall Mean) | |
| 1. In this situation, what proportion of the time do you wear your hearing aid? | XXX | XXX | XXX |
| 2. In this situation, how much does your hearing aid help you? | XXX | XXX | XXX |
| 3. In this situation, with your hearing aid, how much difficulty do you now have? | XXX | XXX | XXX |
| 4. For this situation, how satisfied are you with your hearing aid? | XXX | XXX | XXX |
| | 3M Choice: | 3M Choice: | P-Value |
| 3-6 Months | Unilateral | Bilateral | |
| 1. In this situation, what proportion of the time do you wear your hearing aid? | XXX | XXX | XXX |
| 2. In this situation, how much does your hearing aid help you? | XXX | XXX | XXX |
| 3. In this situation, with your hearing aid, how much difficulty do you now have? | XXX | XXX | XXX |
| 4. For this situation, how satisfied are you with your hearing aid? | XXX | XXX | XXX |

# 4.3 Aim: compare EMA surveys between the two arms in the period between baseline and 3 months, and between 3M choice groups between 3 months and 6 months

For question X, we want to look at the answers to all question X's within a given scenario for the 4 standard scenarios.

Analysis: This will be descriptive. We will use boxplots, violin plots, or another type of plot to describe these scenarios. For each of the 4 standard scenarios, we will display the distributions of the answers to each of the 4 questions for both unilateral and bilateral hearing aid groups (i.e., 1 plot per question with two boxes per scenario for each of the 4 scenario/treatment combos).

Examples of what boxplots and violin plots look like (violin plots can be more informative about the distribution of data because they show the density as well):





## **5 Future Plans**

There are additional items we may wish to explore in the future, at which point a new SAP will be developed. In particular, we may explore EMA responses for the 2 user-nominated scenarios or all 6 scenarios.

# Statistical Analysis Plan (SAP) - Hearing Aid Choice and Switching

**Project:** Evaluation of Unilateral vs Bilateral Hearing Aids for the Treatment of Age-related Hearing Loss **IRB Number:** Pro00106077 Investigator(s): Sherri Smith, AuD, PhD Biostatisticians: **Original Creation Date: 11.16.2023** Version Date: 11.26.2024 ☐ All statistical analyses included in an abstract or manuscript should **Investigator Agreement** reflect the work of the biostatistician(s) listed on this SAP. No changes or additional analyses should be made to the results or findings without discussing with the project biostatistician(s). ☐ All biostatisticians on this SAP should be given sufficient time to review the full presentation, abstract, manuscript, or grant and be included as co-authors on any abstract or manuscript resulting from the analyses. ☐ If substantial additional analysis is necessary or the aims of the project change, a new SAP will need to be developed. ☐ Publications resulting from this SAP are supported in part by the Duke CTSA and must cite grant number UL1TR002553 and be submitted to PubMed Central. □ I have reviewed the SAP and understand that any changes must be documented. Acknowledged by: Click or tap here to enter text. Date: Click or tap to enter a date. **Activity Log** 11.16.2023 Created SAP for outcomes related to hearing aid choice and switching 06.03.2024 Added additional variables, moved questions related to data collected after 3 months to the Future Plans section 07.11.2024 Resolved some comments, added details about potential covariates 07.25.2024 Moved 6-month APHAB into this SAP 10.02.2024 Resolved some comments after discussion (see previous SAP for more details), updated variable names/descriptions 11.26.2024 Resolved some comments after discussion, revised model for identifying associations between baseline covariates and 3M switching or 6M final choice Abbreviated Profile of Hearing Aid Benefit **Acronyms** APHAB **EMA Ecological Momentary Assessment GHABP** Glasgow Hearing Aid Benefit Profile IOI-HA International Outcomes Inventory for Hearing Aids

| SADL | Satisfaction with Amplification in Daily Life |
|------|-----------------------------------------------|
| SSQ | Speech Spatial Qualities |
| HHIE | Hearing Handicap Inventory for Elderly |

## 1 Study Overview

Background/Introduction: The overall goal of the project is to determine the benefit of unilateral or bilateral hearing aid fittings in adults with mild-to-moderate age-related hearing loss. This will address the lack of high-quality evidence supporting bilateral hearing aids over unilateral hearing aids. This project will use a randomized controlled trial with two treatment arms: a bilateral hearing aid fitting group and a unilateral hearing aid fitting group.

#### 1.1 Hearing Aid Switching Aims

- Explore if treatment assignment influences switching configuration at 3 months
- Explore what predicts switching at 3 months
- Describe patient characteristics for switchers vs. non-switchers
- Describe APHAB data (subscales and global score) over time within subgroups of individuals

# 2 Study Population

#### 2.1 Inclusion Criteria

- 50+ years of age
- Mild to moderate, symmetrical SNHL (symmetrical: < 20 dB between ears on average from 500-4000 Hz)
- Open-mindedness to unilateral or bilateral amplification
- No prior hearing aid experience
- Adequate literacy to complete questionnaires
- Willing to purchase study-specific hearing aid(s)

#### 2.2 Exclusion Criteria

- Concerns for middle ear pathology
- Concerns for retrocochlear pathology
- Severe tinnitus as the reason for seeking amplification
- Co-morbid condition that would interfere with study (e.g., dementia, blindness, neurologic pathology)
- History of fluctuating hearing loss

#### 2.3 Data Acquisition

Fill in all relevant information:

| Study design | Randomized controlled trial with 2 arms (bilateral hearing aid, unilateral hearing aid) |
|---|---|
| | Note: Randomization was stratified by clinical site. |
| Data source/how the data were collected | Screening information pulled from EHR data |
| | Baseline surveys captured via in-person interview and |
| | recorded in REDCap |

| Contact information for team member | All data access is through |
|---|---|
| responsible for data | . Questions on data validity |
| collection/acquisition | will go to PI: Sherri Smith (Sherri.smith@duke.edu) |
| Date or version (if downloaded, provide | 10.17.2024 |
| date) | |
| Data transfer method and date | Direct data extraction from REDCap |
| Where dataset is stored | REDCap |
| | Extracted data and analytic datasets are stored on a secure drive in the CRU folder: \\duhs-vclin- nc1\dusom biostats fs\Data\BiostatsCore\CRU\Head and Neck\Smith\PCORI Pro00106077\Data pulls |

Notes:

Description: [insert]

# 3 Outcomes, Exposures, and Additional Variables of Interest

# 3.1 Outcome(s)

| Outcome | Description | Variables and Source | Specifications |
|---|---|---|---|
| Switch configuration at 3 months | Patients are given the opportunity to switch configurations at 3 months. | ha_switch_3m | Binary: 1: Switched configuration 0: Didn't switch Switched configuration is defined as unilateral to bilateral or vice versa (do not count switching unilateral to a different ear as a switch) Switched configuration also includes switching from 1 or 2 to 0 |
| APHAB Global<br>Score | Global<br>communication<br>score at<br>baseline, 3<br>months, 6<br>months | aphab_global_base<br>aphab_global_3m<br>aphab_global_6m | Rescore variables and multiply by 100 1 = 0.99 2 = 0.87 3 = 0.75 4 = 0.50 5 = 0.25 6 = 0.12 7 = 0.01 Reverse score questions 1, 9, 11, 16, 19, 21 |

| | | | Global score: mean of variables in the EC, BN, RV subscale scores (excludes questions 3, 8, 13, 17, 20, 22) |
|---|---|---|---|
| | | | Also potentially used in |
| | | | other models as a covariate |
| APHAB – 4 | EC, BN, RV, AV | aphab_ec_base | Rescore variables and |
| subscales | scales at | aphab_ec_3m | multiply by 100 |
| | baseline, 3 | aphab_ec_6m | • 1 = 0.99 |
| | months, 6 | | • 2 = 0.87 |
| | months | aphab_bn_base | • 3 = 0.75 |
| | | aphab_bn_3m | • 4 = 0.50 |
| | | aphab_bn_6m | • 5 = 0.25 |
| | | | • 6 = 0.12 |
| | | aphab_rv_base | • 7 = 0.01 |
| | | aphab_rv_3m | Reverse score questions 1, |
| | | aphab_rv_6m | 9, 11, 16, 19, 21 |
| | | aphab_av_base | EC: mean of questions 4, |
| | | aphab_av_3m<br>aphab_av_6m | 10, 12, 14, 15, 23 |
| | | | BN: mean of questions 1, 6, |
| | | | 7, 16, 19, 24 |
| | | | RV: mean of questions 2, 5, 9, 11, 18, 21 |
| | | | AV: mean of questions 3, 8, 13, 17, 20, 22 |
| | | | Also potentially used in |
| | | | prediction models as |
| | | | covariates |

# 3.2 Additional Variables of Interest

| Variable | Description | Variables and Source | Specifications |
|----------------|---------------|----------------------|----------------|
| Randomization | hearing aid | assign | Binary |
| assignment | assignment | | 1: unilateral |
| | | | 2: bilateral |
| Clinical site | Which site - | which_site | Binary |
| | Duke or | | 1: Vanderbilt |
| | Vanderbilt? | Character version: | 2: Duke |
| | | which_site_ch | |
| 3 month chosen | Hearing aid | ha_config_3m | Categorical |
| treatment | configuration | | • Right |
| | at 3 months | | • Left |
| | | | • Both |

| | 1 | 1 | T |
|---|---|---|---|
| | | | <ul><li>None</li><li>Missing</li></ul> |
| Gender | | gender | Categorical |
| | | Character version: gender_ch | <ul><li>1: male</li><li>2: female</li></ul> |
| | | 0.11 | • 3: other |
| | | | 99: declined |
| Age | Age at baseline | age_base | Continuous |
| | (years) | Baseline visit is baseline_date | Years from |
| | | _ | baseline_date to dob |
| | | | Baseline visit is |
| | | | defined as |
| | | | aphab_base_date if |
| | | | non-missing, |
| | | | otherwise use |
| _ | | | date_moca |
| Race | | race | Categorical |
| | | Character and a second | 1: African American / Plack |
| | | Character version: race_ch | American/Black • 2: White/Caucasian |
| | | | • 3: Asian |
| | | | 4: Native |
| | | | American/Alaska |
| | | | Native |
| | | | • 5: Native |
| | | | Hawaiian/Pacific |
| | | | Islander |
| | | | 6: More than one |
| | | | race |
| | | | 99: Declined |
| | | | If cell counts are less |
| | | | than 10 for a given |
| | | | category, we will not |
| | | | report the exact cell |
| | | | count. |
| | | | NIH racial categories: |
| | | | -American |
| | | | Indian/Alaska Native |
| | | | -Asian or Asian |
| | | | American |
| | | | -Black or African |
| | | | American |
| | | | -Native |
| | | | Hawaiian/Pacific |
| | | | Islander |
| | | 1 | -White |
| Ethnicity | | ethnicity | Categorical |
| | | | 1: Hispanic or Latino |

| | | Character version:<br>ethnicity_ch | <ul> <li>2: Not Hispanic or<br/>Latino</li> <li>999: Declined</li> <li>If cell counts are less<br/>than 10 for a given<br/>category, we will not<br/>report the exact cell</li> </ul> |
|---|---|---|---|
| Income | Personal<br>Income Last<br>Year | income Character version: income_ch | count. Categorical 0:\$0 1:\$1 to \$9999 2:\$10,000 to \$24,999 3:\$25,000 to \$49,999 4:\$50,000 to \$74,999 5:\$75,000 to \$99,999 6:\$100,000 to \$149,999 7:\$150,000 or greater 999: Prefer not to answer |
| Hearing Aid<br>Health Insurance<br>Benefits | | benefits Character version: benefits_ch | Categorical O: No 1: Yes 998: Not Sure |
| Marital Status | | marital Character version: marital_ch | Categorical 1: married 2: widowed 3: divorced 4: separated 5: never married 999: prefer not to answer |
| Living arrangements | | living Character version: living_ch | Categorical 1: alone 2: with spouse 3: with spouse and others 888: other 999: prefer not to answer |
| Education | | education Character version: education_ch | Categorical 1: less than high school 2: high school 3: some college 4: 4-year degree |

| | | | <ul><li>5: graduate degree</li><li>888: other</li><li>999: prefer not to<br/>answer</li></ul> |
|---|---|---|---|
| Baseline Date<br>Quarter | | baseline_quarter | Categorical |
| Quarter | | | Put baseline date into quarters |
| Cognition<br>(Screened via | Adjusted<br>MoCA score | total_moca | Continuous, 0-30 |
| MoCA) | | | moca31 is a modifier for high school education |
| | | | If moca31=0, then<br>total moca score is the<br>sum of moca1 through<br>moca30 |
| | | | If moca31=1, then total moca score is the minimum of 30 and the sum of moca1 through moca 31 |
| Degree of<br>Hearing Loss – | PTA in better ear | Right ear: pta_right | We will use the pure tone average in the |
| Pure Tone<br>Average | | Left ear: pta_left | better ear. |
| | | Better ear: pta_better | Take the average at frequencies 500, 1000, 2000, 4000 in both ears. The lower average is the better ear. |
| Hearing loss classification | | hearing_loss_class | <ul><li>Mild: pta_better</li><li>&lt;= 40</li><li>Moderate</li><li>pta_better &gt; 40</li></ul> |
| APHAB Change<br>Score | Difference in aided APHAB scores at month 3 and unaided scores at baseline | aphab_change | Scale score – will need to calculate global communication scores at baseline (unaided) and 3 months (aided), subtract (3 months – baseline) A lower score on APHAB is better. |

| APHAB change | Responders vs | Decrease of 25 units: use | Patients with a |
|---|---|---|---|
| score – binary, 3 | non- | aphab_change_responder | decrease of at least 25 |
| months | responders | | units (or 15 units for |
| | for primary | Decrease of 15 units: use | the sensitivity analysis) |
| | APHAB | aphab_change_responder | on the APHAB scale at |
| | outcome | _15 | month 3 will be |
| | | | considered |
| | | | "responders." Patients |
| | | | not returning or who |
| | | | do not have a score at |
| | | | 3 months will be |
| | | | considered "non- |
| | | | responders." |
| | | | Binary (25 unit |
| | | | decrease): |
| | | | • 1 if |
| | | | aphab_change<br><=-25 |
| | | | • 0 else |
| | | | Binary (15 unit |
| | | | decrease); |
| | | | • 1 if |
| | | | aphab_change |
| | | | <=-15 |
| | | | • 0 else |
| IOI-HA | This is | Total score: ioiha_total_3m | Total score: sum |
| | measured | | responses to questions |
| | only at 3 and | | 1-7 (should be on a |
| | 6 months | | range between 1-5). |
| | | | Item 8 is self- |
| | | | perceived hearing |
| | | | difficulty used for |
| | | | normative purposes |
| | | | (currently not used as |
| | | | part of total score) |
| | | | This is initially coded |
| | | | as 0 to 4 in REDCap – |
| | | | changed to 1-5 |
| | | | Currently, we're |
| | | | treating IOI-HA total |
| | | | score as continuous, |
| | | | but this may need to |
| | | | be treated as ordinal. |
| | | | Higher scores are |
| | | | better |

| SADL | This is | Global score: sadl_global_3m | Questions 1 – 15 are |
|---|---|---|---|
| | measured | Danii a affaal a baaala | used. This is scored |
| | only at 3 and | Positive effect subscale: | from 1-7 (or reversed |
| | 6 months. | sadl_positive_effect_3m | for questions 2, 4, 7,<br>13). |
| | Note: the | Service cost subscale: | - / |
| | "sister" | sadl_service_cost_3m | There are 4 subscales: |
| | questionnaire | | Positive Effect, Service |
| | at baseline is | Negative features subscale: | & Cost, Negative |
| | ECHO | sadl_negative_features_3m | Features, Personal |
| | | | Image. For each |
| | | Personal image subscale: | subscale, the average |
| | | sadl_personal_image_3m | score is calculated. |
| | | | For the global score, |
| | | | this is the mean of the |
| | | | scores for all items |
| | | | (excluding questions |
| | | | 11 and 14 if |
| | | | applicable). |
| | | | Higher scores are |
| | | | better (higher |
| | | | satisfaction). |
| | | | See PCORI Scoring file |
| | | | for more details |
| SSQ | This is | Change score: ssq_change | 3 subscales: Speech is |
| | measured at | | questions 1 – 14 |
| | baseline, 3 | Baseline: | (corresponds to the |
| | months, and 6 | Overall score: | "pt1" variables). |
| | months | ssq_overall_base | Spatial is 17 questions |
| | | | (corresponds to the |
| | | Speech/hearing subscale: | "pt2" variables). |
| | | ssq_speech_hearing_base | Qualities is 18 |
| | | Spatial/hearing subscale: | questions (correspond to the "pt3" variables). |
| | | ssq_spatial_hearing_base | to the pts variables). |
| | | | Overall score: mean of |
| | | Qualities of hearing subscale: | the items. |
| | | ssq_qualities_of_hearing_base | |
| | | | For instances where |
| | | 3-Months: | people mark NA and a |
| | | Overall score: ssq_overall_3m | value, if the value is |
| | | Connected the second second | 50, set as NA. If a |
| | | Speech/hearing subscale: | value other than 50, |
| | | ssq_speech_hearing_3m | use that value. |
| | | Spatial/hearing subscale: | We will also create a |
| | | Spatial/hearing subscale: ssq_spatial_hearing_3m | We will also create a change score as the difference in the |

| | | Qualities of hearing subscale: | overall score between |
|---|---|---|---|
| | | ssq_qualities_of_hearing_3m | 3 months and baseline |
| | | | (3 months – baseline) |
| | | | Higher scores are better |
| HHI-E | This is measured at | Change score: hhie_change | Yes = 4 points,<br>Sometimes = 2 points, |
| | baseline, 3 months, and 6 | Baseline: Total score: hhie total base | and No = 0 points. |
| | months | | Total scale score = |
| | | Situational subscale: | sum of all 25 items |
| | | hhie_situational_base | Situational subscale: |
| | | Emotional subscale: | questions 1, 3, 6, 8, |
| | | hhie_emotional_base | 10, 11 13, 15, 16, 19,<br>21, 23 |
| | | 3-Months: | · |
| | | Total score: hhie_total_3m | Emotional subscale: questions 2, 4, 5, 7, 9, |
| | | Situational subscale: | 12, 14, 17, 18, 20, 22, |
| | | hhie_situational_3m | 24, 25 |
| | | Emotional subscale: | We will also create a |
| | | hhie_emotional_3m | change score as the |
| | | | difference in the total scale score between 3 |
| | | | months and baseline |
| | | | (3 months – baseline) |
| | | | Lower scores are better |
| Hours of Hearing | Multiple time | Right ear: | How many hours on |
| Aid Use | periods (every scheduled | r_avg_hrs_3m<br>r_avg_hrs_3m_na (if right HA | average the right/left HA was worn. |
| | visit and | is NA) | TIA Was Worth. |
| | unscheduled | | NA variables: value of |
| | follow ups) | Left ear: I_avg_hrs_3m | 1 if that HA was NA |
| | | _avg_hrs_3m_na | |
| GHABP Unaided | GHABP is | Question 2 average, 4 | For questions 2 and 3 |
| S Characa | measured at | standard scenarios: | (IF they answer yes to |
| | baseline | ghabp_q2_4block_base | question 1), doing this |
| | (unaided) | Ouestion 2 average 4 | separately by |
| | | Question 3 average, 4 standard scenarios: | question: |
| | | ghabp_q3_4block_base | 1. Subtract 1, |
| | | | multiply by 25, |

| | | | average answer to question across 4 standard scenarios There are 6 scenarios (4 standard, 2 user- nominated) Note that question 1 |
|---|---|---|---|
| | | | just asks if this<br>scenario has<br>happened —<br>participants are only<br>included in the<br>averages if they<br>answer "yes" |
| | | | Lower scores are better for both questions |
| GHABP Aided | GHABP is<br>measured at 3<br>months<br>(aided) | Question 2 average, 4 standard scenarios: ghabp_q2_4block_3m Question 3 average, 4 standard scenarios: ghabp_q3_4block_3m Question 4 average, 4 standard scenarios: ghabp_q4_4block_3m | For questions 3-6 (IF they answer yes to question 1), doing this separately by question: 1. Subtract 1, multiply by 25, average answer to question across 4 standard scenarios |
| | | Question 5 average, 4 standard scenarios: ghabp_q5_4block_3m Question 6 average, 4 standard scenarios: ghabp_q6_4block_3m | Note: ignore current question 2 for analyses as it is nonstandard but report on this in a descriptive table There are 6 scenarios (4 standard, 2 usernominated) |
| | | | Note that question 1 just asks if this scenario has happened – participants are only included in the |

| | | | averages if they answer "yes" Higher/lower scores are better depending |
|---|---|---|---|
| | | | on question |
| Binaural<br>loudness<br>summation | CSL level right CSL level left CSL level both | binaural_r_base<br>binaural_l_base<br>binaural_both_base | Continuous |
| Dichotic digit test | Right ear directed Left ear directed Free recall both ears Right ear free recall Left ear free recall | dichotic_r_base<br>dichotic_l_base<br>dichotic_free_both_base<br>dichotic_free_r_base<br>dichotic_free_l_base | Continuous |
| Speech and<br>Noise Test | Baseline (unaided) and 3-months (aided) Speech and noise 0 degrees (collocated) Speech left, noise right Noise left, speech right | Baseline: sin_collocated_base sin_right_base sin_left_base 3-Months: sin_collocated_3m sin_right_3m sin_left_3m Change: sin_collocated_change sin_r_change sin_r_change May also want change scores for speech to aided side and speech to unaided side | Change scores: 3m-baseline for each of collocated, speech left/noise right, noise left/speech right Positive values for unaided/aided variables indicate speech is louder than noise; negative indicate speech is under the noise For unilateral assigned, also have speech to aided side (advantage) and speech to unaided side (disadvantage). Speech to aided (advantage): If assigned R, this is noise left, speech |

| | | | If assigned L, this is<br>speech left, noise<br>right |
|---|---|---|---|
| | | | Speech to unaided (disadvantage): If assigned R, this is speech left, noise right If assigned L, this is noise left, speech right |
| | | | Lower scores are better |
| Auditory<br>Working | Unaided and<br>Aided (3 | Change scores: warrm_recog_change | Continuous |
| Memory | months) Recognition, judgement, recall | warrm_recall_change Baseline: warrm_recog_base warrm_recall_base | Sum questions 2-6 for each tasks (recognition, judgement, recall) separately and get a % |
| | recan | warrm_judge_base | correct (out of 20) |
| | | 3-Months: warrm_recog_3m warrm_recall_3m warrm_judge_3m | Construct change scores as difference between 3 months and baseline for recognition and recall. |
| | | | Judgement is more of<br>a sanity check (<90%<br>means they probably<br>aren't engaged) |
| | | | Higher scores are better |
| ЕСНО | Baseline only Note: this is | Global score:<br>echo_global_base | Questions 1 – 15 are used. This is scored from 1-7 (or reversed |
| | the "sister" questionnaire to SADL | Positive effect subscale: echo_positive_effect_base | for questions 2, 4, 7, 13). |
| | (aided) | Service cost subscale: echo_service_cost_base | There are 4 subscales: Positive Effect, Service & Cost, Negative |
| | | Negative features subscale: echo_negative_features_base | Features, Personal<br>Image. For each<br>subscale, the average |
| | | Personal image subscale: echo_personal_image_base | score is calculated. |

| 53 | 33 | For the global score, |
|----|----|-------------------------|
| | | this is the mean of the |
| | | scores for all items |
| | | (excluding question 11 |
| | | if applicable). |
| | | Higher scores are |
| | | better (higher |
| | | expectations). |
| | | See PCORI Scoring file |
| | | for more details |

# 4 Statistical Analysis Plan

Analysis: To be completed by December 31, 2024.

#### 4.1 Descriptive Table of Switched Configuration Status by Assigned Treatment

Analysis: This will be descriptive. As appropriate, we will present the frequency with percentage (see Table 1). Note that "switched configuration" will be defined as yes for those who switched configuration at 3 months and will be defined as no for those who did not switch configuration at 3 months.

| Table 1: Switched HA Configuration and Choice vs. Assigned Treatment | | | |
|---|---|---|---|
| | Assigned Unilateral Left (N=XXX) | Assigned Unilateral Right (N=XXX) | Assigned Bilatera<br>(N=XXX) |
| Switched Configuration at | | | |
| 3 Months | | | |
| No | XXX (%) | XXX (%) | XXX (%) |
| Yes | XXX (%) | XXX (%) | XXX (%) |
| Missing | XXX (%) | XXX (%) | XXX (%) |
| Hearing Aid Configuration | | | |
| Choice at 3 Months | | | |
| Unilateral Left | XXX (%) | XXX (%) | XXX (%) |
| Unilateral Right | XXX (%) | XXX (%) | XXX (%) |
| Bilateral | XXX (%) | XXX (%) | XXX (%) |
| None | XXX (%) | XXX (%) | XXX (%) |
| Missing | XXX (%) | XXX (%) | XXX (%) |

#### 4.2 Investigate if assigned treatment influences switching at 3 months

Analysis: This will be done using assigned treatment for patients who have information on switching status at 3 months. This analysis will be performed using logistic regression where the outcome is switching status (the probability modelled is switching). The only covariate included in this model will be assigned treatment. A similar model will be fit for the binary outcome 6M HA configuration choice (unilateral vs bilateral).

Hearing Aid Switching Status =  $\beta_0 + \beta_1 * treatment$  assignment

| Table 2 Logistic Regression OR Estimate Probability Modelled: Switched | | | |
|---|---|---|---|
| Covariate | OR | 95% C.I. | P-Value* |
| Hearing Aid Assignment (Reference:<br>Bilateral) | | | |
| Unilateral | XXX | (XXX, XXX) | XXX |

#### 4.3 Investigate what predicts switching at 3 months

Analysis: This will be done for all randomized patients who are not missing scores or other predictors of interest. This analysis will be performed using the LASSO for logistic regression where the outcome is switching status (the probability modelled is switching) or 6M HA configuration choice (modelled probability is unilateral). Covariates (denoted generally as L below) to include in these models are age at baseline, gender, pure tone average in the better ear, baseline global HHI-E, baseline APHAB Global, baseline APHAB AV, binaural loudness summation (both), REAfree (Dichotic Digits, free right minus free left), REAdirect (Dichotic Digits, direct right minus direct left), cognitive effect LE (Dichotic Digits, direct left minus free left), cognitive effect RE (Dichotic Digits, direct right minus free right), AWARRM recall, and education-adjusted MoCA total score. The selected variables, their odds ratios, and 95% confidence intervals constructed from post-selection inference methods (R package 'selectiveInference') will be reported.

Hearing Aid Switching Status =  $\beta_0 + \beta_L * L$ 

| Table 3: Logistic Regression OR Estimates Probability Modelled: Switched HA Configuration | | |
|---|---|---|
| Covariate | OR | P-S 95% C.I. |
| Covariate 1 (Ref: category) | | |
| Category x | XXX | (XXX, XXX) |
| Covariate 2 | XXX | (XXX, XXX) |

#### 4.4 Describe patient characteristics for those who switch their HA configuration vs. those who don't

Analysis: The characteristics from "non-switchers" will be compared to "switchers" with the use of a "Table 1". As appropriate, we will present the mean with standard deviation (SD), median with interquartile range (IQR), and ranges (min and max), or frequency with percentage. A similar table will be constructed with participants stratified by 6M HA configuration choice.

| | Non-Switchers (N=XXX) | Switchers (N=XXX) |
|-----------------------|-----------------------|-------------------|
| Clinical Site | | |
| Duke | XXX (%) | XXX (%) |
| Vanderbilt | XXX (%) | XXX (%) |
| Gender | | |
| Female | XXX (%) | XXX (%) |
| Male | XXX (%) | XXX (%) |
| Other | XXX (%) | XXX (%) |
| Age at Baseline Visit | | |
| N | XXX | XXX |

| Missing | XXX | XXX |
|---------------------------------------|-----------|-----------|
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX , XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX |
| Race | | |
| American Indian/Alaska Native | XXX (%) | XXX (%) |
| Asian | XXX (%) | XXX (%) |
| Black or African American | XXX (%) | XXX (%) |
| White | XXX (%) | XXX (%) |
| More than one race | XXX (%) | XXX (%) |
| Native Hawaiian/Pacific Islander | XXX (%) | XXX (%) |
| Declined | XXX (%) | XXX (%) |
| Ethnicity | | |
| Hispanic or Latino | XXX (%) | XXX (%) |
| Not Hispanic or Latino | XXX (%) | XXX (%) |
| Declined | XXX (%) | XXX (%) |
| Personal Income Last Year | | |
| \$0 | XXX (%) | XXX (%) |
| \$1 to \$9999 | XXX (%) | XXX (%) |
| \$10,000 to \$24,999 | XXX (%) | XXX (%) |
| \$25,000 to \$49,999 | XXX (%) | XXX (%) |
| \$50,000 to \$74,999 | XXX (%) | XXX (%) |
| \$75,000 to \$99,999 | XXX (%) | XXX (%) |
| \$100,000 to \$149,999 | XXX (%) | XXX (%) |
| \$150,000 or greater | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) |
| Hearing Aid Health Insurance Benefits | | |
| No | XXX (%) | XXX (%) |
| Yes | XXX (%) | XXX (%) |
| Not sure | XXX (%) | XXX (%) |
| Marital Status | | |
| Married | XXX (%) | XXX (%) |
| Widowed | XXX (%) | XXX (%) |
| Divorced | XXX (%) | XXX (%) |
| Separated | XXX (%) | XXX (%) |
| Never married | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) |
| Living Arrangements | | |
| Alone | XXX (%) | XXX (%) |
| With spouse | XXX (%) | XXX (%) |
| With spouse and others | XXX (%) | XXX (%) |
| Other | XXX (%) | XXX (%) |
| Prefer not to answer | XXX (%) | XXX (%) |

| Education | | |
|-------------------------------------------|-----------|-----------|
| Less than high school | XXX (%) | XXX (%) |
| High school | XXX (%) | XXX (%) |
| Some college | XXX (%) | XXX (%) |
| 4-year degree | XXX (%) | XXX (%) |
| Graduate degree | XXX (%) | XXX (%) |
| Other | XXX (%) | XXX (%) |
| Quarter of Baseline Visit | | |
| 2021 Q2 | XXX (%) | XXX (%) |
| 2021 Q3 | XXX (%) | XXX (%) |
| | XXX (%) | XXX (%) |
| Total MoCA Score | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX , XXX | XXX , XXX |
| Range | XXX - XXX | XXX - XXX |
| Pure Tone Average in Better Ear | | |
| N | XXX | XXX |
| Missing | XXX | XXX |
| Mean (SD) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX |
| Q1, Q3 | XXX,XXX | XXX,XXX |
| Range | XXX - XXX | XXX - XXX |
| Hearing Loss Classification in Better Ear | | |
| Mild | XXX (%) | XXX (%) |
| Moderate | XXX (%) | XXX (%) |

#### 4.5 Describe APHAB data over time

**Analysis:** This will be done graphically. We will plot the average APHAB subscale scores and global score over time (baseline, 3-months, 6-months). These plots will be grouped by hearing aid assignment/choice such as: individuals assigned 1 hearing aid and kept 1 hearing aid, individuals assigned 2 hearing aids and kept 2 hearing aids, and individuals who switched hearing aid configuration at 3 months. We may explore additional groups depending on the patterns we see.

We will use these plots to describe general trends (i.e., describe if score trajectories seem to differ by hearing aid configuration group).

#### 5 Future Plans

There are additional items we may wish to explore in the future, at which point a new SAP will be developed, related to 6-month outcomes and/or switching at the 6-month time point.